Title: OPEN-LABELED TRIAL OF DIRECT-ACTING ANTIVIRAL TREATMENT OF HEPATITIS C NEGATIVE PATIENTS WHO RECEIVE KIDNEY TRANSPLANTS FROM HEPATITIS C POSITIVE DONORS (THINKER)

**Study Identifier: NCT02743897** 

Date: October 1, 2020, PROTOCOL V6.0

# OPEN-LABELED TRIAL OF DIRECT-ACTING ANTIVIRAL TREATMENT OF HEPATITIS C NEGATIVE PATIENTS WHO RECEIVE KIDNEY TRANSPLANTS FROM HEPATITIS C POSITIVE DONORS (THINKER)

Test drug: Zepatier or another antiviral regimen for hepatitis C virus infection

Clinical study phase: II

Sponsor: N/A

Funder: Merck

IND# Exempt

IRB# **823833** 

NCT# **NCT02743897** 

Stacey Prenner, MD

Perelman School of Medicine at the University of Pennsylvania

Co-principal

215-760-0307

Investigators: Peter Reese, MD, MSCE

Perelman School of Medicine at the University of Pennsylvania

215-900-3782

The study will be conducted in adherence with the protocol, ICH-GCP and any applicable regulatory requirements.

#### Confidential

The information provided in this document is strictly confidential and is intended solely for the guidance of the clinical investigation. Reproduction or disclosure of this document - whether in part or in full - to parties not associated with the clinical investigation, or its use for any other purpose, without the prior written consent of the principal investigator is not permitted.

Throughout this document, symbols indicating proprietary names (®, tm) are not displayed. Hence, the appearance of product names without these symbols does not imply that these names are not protected.

### 1 SYNOPSIS

| Title | Open-Labeled Trial Of Direct-Acting Antiviral Treatment Of Hepatitis C-Negative Patients Who Receive Kidney Transplants From Hepatitis C-Positive Donors |
|---|---|
| Clinical study phase | II |
| Study objectives | This study is being conducted to determine safety and efficacy of transplanting kidneys from HCV virus (HCV)-infected donors into HCV-negative patients on the kidney transplant waitlist, who will then be treated with Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment status post-single kidney transplantation. |
| | Primary aim: 1. Primary efficacy objective: to determine sustained virologic response (SVR) rates of open-label Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment in HCV-negative patients who receive a kidney transplant from an HCV-infected donor, leading to post-transplantation de-novo HCV infection. |
| | 2. <u>Primary safety objective</u> : to determine the safety of administration of open-<br>label Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment<br>among HCV-negative patients who receive a kidney transplant from an<br>HCV-infected donor and develop post-transplant HCV infection. |
| | Secondary aims: |
| | 3. To determine 1-year graft survival rates of HCV-negative kidney transplant patients who receive a kidney transplant from an HCV-infected donor, including those who spontaneously clear HCV (and those who receive openlabel Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment upon development of de-novo HCV. |
| | 4. To evaluate rates of spontaneous clearance of HCV among HCV-negative patients who receive a single kidney transplant from an HCV-infected donor. |
| Indication | Chronic HCV post-kidney transplantation |
| Diagnosis and main criteria for inclusion | <ul> <li>Inclusion criteria</li> <li>Must be waitlisted for a kidney transplant</li> <li>Listed for an isolated kidney transplant with ≤2555 days of accrued transplant waiting time and/or ≤2555 days of dialysis time for blood group A, B, or O, by enrollment</li> <li>Listed for an isolated kidney transplant with ≤1825 days of accrued transplant waiting time and/or ≤1825 days of dialysis time for blood group AB, by enrollment</li> <li>No available living kidney donor</li> <li>Between 30-70 years of age, by enrollment</li> <li>Have a panel reactive antibody level ≤97%</li> </ul> |

- eGFR <15ml/min/1.73m<sup>2</sup> as calculated using the 4 variable MDRD equation
- Obtained agreement for participation from the patient's treating transplant nephrologist
- Able to travel to the University of Pennsylvania for routine post-transplant visits and study visits for a minimum of 6 months after transplantation
- Women must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) following transplant due to the increased risk of birth defects and/or miscarriage
- Both men and women must agree to use at least one barrier method to prevent any secretion exchange
- No active illicit substance abuse
- Weigh at least 50kg
- Inclusion criteria for treatment (not for entry as study patient) will include any detectable HCV RNA level
- Able to provide informed consent

#### Exclusion criteria

- Hepatocellular carcinoma
- Patients with primary focal segmental glomerulosclerosis (FSGS), FSGS
  recurring after previous transplant, or disease process with increased risk of
  causing early graft failure as assessed by the transplant nephrologist and/or
  the investigator team
- HIV positive
- HCV RNA positive (can be isolated HCV antibody positive provided the subject has no history of previously treated HCV)
- Hepatitis B surface antigen positive
- Any other chronic liver disease (excluding non-alcoholic fatty liver disease (NAFLD) with abnormal liver enzymes
- Persistently elevated liver transaminases
- Significant hepatic fibrosis on screening elastography (≥F2 fibrosis)
- Pregnant or nursing (lactating) women
- Known allergy or intolerance to tacrolimus that would require post-transplant administration of cyclosporine, rather than tacrolimus given the drug-drug interaction between cyclosporine and certain direct-acting antivirals (DAA)
- Waitlisted for a multi-organ transplant (e.g., pancreas-kidney, heart-kidney, etc.)
- Significant cardiomyopathy (e.g., left-ventricular heart failure, pulmonary hypertension).

#### Study design

Open-labelled pilot clinical trial of Zepatier (MK-5172 and MK-8742/Grazoprevir + Elbasvir), Mavyret, Epclusa, or another appropriate antiviral treatment in HCV-negative subjects with end-stage renal disease receiving a kidney transplant from a HCV-positive donor. Eligible subjects will receive a kidney transplant from a deceased-donor with detectable HCV nucleic acid, and then will receive Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment after kidney transplantation when infection with HCV is confirmed in these kidney transplant recipients. For Zepatier,

| | treatment will be complete after 12 weeks.* For Mavyret treatment will be complete after 8 weeks, and Epclusa treatment will be complete after 12 weeks. * Patients with Genotype 1a and Genotype 1 with an unknown subtype will have baseline NS5A drug resistance assay testing checked at the start of treatment, and if patients have polymorphisms at positions M28, Q30, L31, and/or Y93, treatment with Zepatier will be extended to 16 weeks, rather than 12 weeks, and renally-adjusted Ribavirin at the clinician's discretion will be initiated, and continued for the remainder of therapy (until the 16 week mark). Such a strategy will provide optimal treatment, without delaying therapy prior to receipt of results of NS5A drug resistant testing. |
|---|---|
| Study observations | <ul> <li>Laboratory tests including hepatic function panel at baseline and at multiple time points during follow-up.</li> <li>Fibroscan at screening, post-transplant (prior to treating HCV), and post-treatment</li> <li>HCV RNA prior to treatment, on treatment, and 4 and 12 weeks after completing Zepatier.</li> </ul> |
| Type of control | None |
| Number of subjects | Estimated 75 HCV-negative subjects transplanted with a kidney from an HCV-positive donor |
| Plan for statistical analysis | <ul> <li>Primary endpoint: <ul> <li>Post-treatment sustained virologic response (SVR)</li> </ul> </li> <li>Secondary endpoints: <ul> <li>Determine if there are major adverse events attributable to HCV therapy in post-kidney transplant patients.</li> <li>Evaluate 1-year kidney graft survival in HCV-negative patients who receive a kidney transplant from an HCV-positive donor</li> <li>Determine the rates of spontaneous HCV clearance among HCV-negative patients with end-stage renal disease receiving a kidney from an HCV-positive donor</li> </ul> </li> <li>Data analysis: <ul> <li>The primary analysis will be based on a calculation of SVR rates (number of subjects with SVR-12; negative HCV RNA 12 weeks after completing Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment) / (number of subjects treated with Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment post-kidney transplantation)</li> </ul> </li> </ul> |

### 2 TABLE OF CONTENTS

### **TABLE OF CONTENTS**

| 1 | | sis | |
|---|---|---|---|
| 2 | | of contents | |
| 3 | Abstra | rct | 7 |
| 4 | Chapte | er 1: Background And Significance | 8 |
| 4. | 1. | Background | 8 |
| 4. | 2. | Rationale of the study | 9 |
| 4. | 3. | Zepatier for recipients of kidney transplants from donors with genotype 1 or 4 HCV | 9 |
| 5 | Chapte | er 2: Objectives And Specific Aims | 11 |
| 5. | 1. | Objectives | 11 |
| 5. | | Specific aims | |
| 6 | Chapte | er 3: Screening And Subject Selection | 12 |
| 6. | 1. | Recruitment: identification and screening process | 12 |
| 6. | 2. | Subject selection criteria | 13 |
| | 6.2.1. | Inclusion criteria | |
| | 6.2.2. | Exclusion criteria | 13 |
| 6. | 3. | Donor Organ Selection Criteria | 14 |
| | 6.3.1. | Donor Evaluation | 14 |
| | 6.3.2. | Drug Resistance Testing | 15 |
| 7 | Chapte | er 4: Treatments | |
| 7. | 1. | Zepatier (grazoprevir and elbasvir) for kidney recipients with HCV genotype 1 or genotyp | e 4 |
| in | fection | 16 | |
| | 7.1.1. | Administration of Zepatier | |
| | 7.1.2. | Drug logistics and accountability | |
| | 7.1.3. | Destruction and return | 18 |
| | 7.1.4. | Zepatier Initial Treatment Failures | |
| 8 | Chapte | er 5: Data Collection | 20 |
| 8. | 1. | Study visits | 20 |
| | 8.1.1. | Informed consent | 20 |
| | 8.1.2. | Screening | 20 |
| | 8.1.3. | Post-Kidney Transplant | 21 |
| | 8.1.5. | Long-term outcomes and Future research | |
| 8. | 2. | Study schedule of procedures | 27 |
| | 8.2.1. | Visits, lab testing, and other clinical testing | |
| | 8.2.2. | Blood sampling volumes | |
| 8. | 3. | Subject retention and drug adherence | 30 |
| 9 | Chapte | er 6: Assessment Of Efficacy And Outcome Measures | 31 |
| 9. | 1. | Assessments of Efficacy | 31 |
| | 9.1.1. | Sustained Virologic Response (SVR) | 31 |
| 9. | 2. | Secondary Outcome Measures | 31 |
| | 9.2.1. | Safety | 31 |
| | 9.2.2. | Graft Survival | |
| | 9.2.3. | Spontaneous Clearance or Non-Transmission of HCV | 31 |
| 10 | Chapte | er 7: Statistical Considerations | 32 |

| - | 10.1. | Study Design | 32 |
|---|---|---|---|
| - | 10.2. | Disposition of Subjects and Baseline Comparisons | 32 |
| • | 10.3. | Analyses of Outcome Measures | 32 |
| : | 10.4. | Missing Data and Dropouts | 32 |
| • | 10.5. | Protocol Violations | 32 |
| : | 10.6. | Safety Analysis | 32 |
| 11 | Chaptei | 8: Quality Control and Data Handling | .33 |
| : | 11.1. | Personnel Training | 33 |
| : | 11.2. | Data Quality | 33 |
| : | 11.3. | Audit and Inspection | 33 |
| : | 11.4. | Archiving | 33 |
| 12 | Chaptei | 9: Participant Safety and Confidentiality | .34 |
| : | 12.1. | Informed Consent and eConsent (i.e., remote consent) | 34 |
| : | 12.2. | Institutional Review Board Process | |
| : | 12.3. | Insurance | 34 |
| : | 12.4. | Laboratory Values | 35 |
| | 12.4.1. | Chemistry | 35 |
| | 12.4.2. | Serum virologic testing | 35 |
| | 12.4.3. | Pregnancy Testing | 35 |
| | 12.4.4. | Hepatitis C Viral Kinetics | |
| | 12.5. | Zepatier Related Laboratory Abnormalities and Drug Interactions | |
| | 12.6. | Mavyret Related Laboratory Abnormalities and Drug Interactions | |
| | 12.7. | Epclusa Related Laboratory Abnormalities and Drug Interactions | |
| | 12.8. | Other Events | |
| | 12.9. | Safety and Adverse Events | 40 |
| | 12.9.1. | Definitions | 40 |
| | 12.9.2. | Classifying Adverse Events | 41 |
| | 12.9.3. | Interpretation of Definitions | |
| | 12.9.4. | Reporting Procedures for Unanticipated Problems, Adverse Events, and Adverse Device Effects | |
| • | 12.10. | Subject Withdrawal | |
| • | 12.11. | Confidentiality of Study Data | 47 |
| | 12.12. | Potential Risks | 48 |
| | 12.12.1 | Risks of Study Procedures | 48 |
| | 12.12.2 | Risk of Genotyping Failure | |
| | 12.12.3 | | |
| | 12.12.4 | - | |
| | 12.12.5 | , | |
| • | 12.13. | Risk of HCV Transmission | |
| - | There is a s | small risk of transmission of HCV from the study subject to intimate partners during sexual activity | у. |
| | | very low and should be reduced even further due to requirements for subjects to use barrier | • |
| | | during sexual activity. | 50 |
| | 12.14. | Potential Benefits | |
| | | Alternatives | |
| | 12.16. | Ethical Considerations | |
| 13 | | · 11: Good Clinical Practice | |
| 14 | • | 12: References | |

### 3 ABSTRACT

The scarcity of organs for kidney transplantation and high death rates on the waiting list have led some patients to accept kidneys with elevated risks of disease transmission, including infection and cancer. In contrast, transplant teams often discard kidneys from donors with HCV because of the many complications caused by HCV infection and historical barriers to successful treatment. However, new antiviral therapies with cure rates of >95% for all HCV genotypes should prompt transplant leaders to view HCV-positive organs as a valuable opportunity both for transplant candidates with chronic HCV and for uninfected patients awaiting transplantation. The resulting expansion of the donor pool has the potential to save hundreds of lives annually. In many regions of the us, average waiting times for kidney transplantation surpass five years, especially for patients with blood types A, B, or O. Current regulations from the United Network for Organ Sharing (UNOS, the organization that oversees the US system of solid organ transplantation) and the Health Resources and Services Administration (HRSA) do not prohibit the use of HCV-positive kidneys for HCV-negative recipients

We will perform an extension of our initial pilot trials to prove feasibility of knowingly using HCV-positive organs for HCV-negative recipients, by transplanting up to 75 HCV-negative subjects with kidneys from HCV-positive donors, and then treating these subjects' with Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment in the early post-transplant phase in order to cure their HCV. If any subjects clear HCV spontaneously within the first four weeks post-transplantation, and do not require treatment, subjects will be added until there have been 75 HCV-negative subjects who receive a kidney transplant from an HCV-positive donor, develop HCV, and are then treated for their HCV with Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment.

### 4 CHAPTER 1: BACKGROUND AND SIGNIFICANCE

#### 4.1. Background

The scarcity of organs for kidney transplantation and high death rates on the waiting list have led some patients to accept kidneys with elevated risks of disease transmission, including infection and cancer. In certain cases, such as the transmission of cytomegalovirus, physicians can anticipate these events and institute preventive measures. In contrast, transplant teams often discard kidneys from donors with HCV because of the many complications caused by HCV infection and historical barriers to successful treatment. However, new antiviral therapies with cure rates of >95% in all HCV genotpyes should prompt transplant leaders to view HCV-positive organs as a valuable opportunity both for transplant candidates with chronic HCV and for uninfected patients awaiting transplantation.<sup>1-5</sup> the resulting expansion of the donor pool has the potential to save hundreds of lives annually. In many regions of the US, average waiting times for kidney transplantation surpass five years, especially for patients with blood types A, B, or O. Average waitlist death rates are 4% per year, and much higher among diabetics and the elderly. The kidney transplant waiting list exceeds 100,000 candidates, while thousands of other dialysis patients who might benefit from transplant are never referred.

This reluctance to use HCV-positive organs reflects in part past experiences with post-transplant HCV complications, both hepatic (e.g., cirrhosis) and extra-hepatic (e.g., glomerulonephritis that can injure the kidney transplant), but largely from low efficacy rates of interferon-based regimens, which also carried a substantial risk of transplant rejection due to interferon. However, new all-oral HCV therapies should change the paradigm by which we utilize organs from HCV-infected donors. <sup>6</sup> Importantly, early evidence suggests that response rates to new HCV therapies in the transplant setting should be as successful as treatment in the non-transplant setting (based on data on liver transplant recipients presented at the 2014 AASLD liver meeting <sup>7</sup> and our own publications in the Annals of Internal Medicine and the American Journal of Transplantation). <sup>8,9</sup>

Current regulations from the United Network for Organ Sharing (UNOS, the organization that oversees the US system of solid organ transplantation) and the Health Resources and Services Administration (HRSA) do not prohibit the use of HCV-positive kidneys for HCV-negative recipients, and it has been done in rare cases for the last 20 years.

Based on national registry data, from 2005-2014, among 3,273 HCV-positive deceased donors (yielding a potential 6,546 kidneys) consented for organ donation, 2,402 (37.0%) of these kidneys were transplanted, while 4,144 (63.0%) were discarded. These discarded HCV-positive kidneys could have led to a lifesaving transplant to 400 kidney patients annually, resulting in 12,000 years of graft-life over a 5-year period. Such an endeavor would be a paradigm shift in the field of solid organ transplantation, and could change the way in which 'high-risk' organs are viewed for transplantation. Importantly, with regards to treatment of these patients and post-transplant renal function, based on published data, approximately 90% of kidney transplant recipients will have an estimated glomerular filtration rate ≥30ml/min/1.73m². However, some patients will not achieve this threshold, and/or will require treatment for their HCV prior to week 6 post–transplant. Thus, treatment of these patients with Zepatier in the setting of genotype 1 or 4 infection is ideal in comparison to other available treatment options for HCV given its optimal profile with regards to treating patients with impaired renal function. Since the release of Zepatier, newer antivirals have been released that are safe to use in individuals with a GFR <30 in phase 3 or real world studies and have been shown to be highly effective in eradicating HCV. These medications include Mavyret and Epclusa.

#### 4.2. Rationale of the study

We will perform an extension of our pilot trials to prove feasibility of knowingly using HCV-infected organs for HCV-negative recipients, by transplanting up to 75 HCV-negative subjects with kidneys from HCV-infected donors, and then treating these subjects' with Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment in the early post-transplant phase in order to cure their HCV.

### 4.3. Zepatier for recipients of kidney transplants from donors with genotype 1 or 4 HCV

Open-label Zepatier (grazoprevir 100 mg and elbasvir 50 mg) will be administered.<sup>3,4</sup> Zepatier is a fixed-dose combination tablet without ribavirin. GZR is an HCV NS3/4a inhibitor while EBR is an HCV NS5A inhibitor. Both grazoprevir and elbasvir are direct-acting antivirals, which together form an effective therapy for HCV and reduce the likelihood and effects of long-term liver-related HCV complications. GZR/EBR exhibits broad in vitro activity against most HCV genotypes and in vitro activity against many clinically relevant RAVs.<sup>3,4</sup>

Zepatier has been evaluated globally in multiple phase I, II, and III trials to treat HCV.<sup>3,4</sup> Randomized, placebocontrolled trials have been carried out, which led to FDA approval for Zepatier as a treatment for genotype 1 or 4 HCV.

As of July 1, 2015, a diverse population of over 1000 HCV patients has been exposed to Zepatier either as a single agent or in combination with ribavirin or sofosbuvir in phase I/II/III studies. Zepatier has been generally well tolerated at doses of 50-100 mg GZR and 50 mg EBR orally once daily. It has been comparably effective across all subgroups it has been tested in, including non-cirrhotic and/or treatment-naïve subjects.<sup>3,4</sup>

Headaches, fatigue, and nausea represent the most common adverse drug reactions with Zepatier.<sup>3,4</sup> Other drug-related adverse events have included arthralgia, insomnia, diarrhea, dizziness, pyrexia, and asthenia.<sup>3,4</sup> Drug-related serious adverse events are uncommon, but include allergic reactions, possible adverse interactions with other medications, or elevated liver enzymes. In past Zepatier trials, the majority of the adverse events were reversible. These adverse events are usually grade 1 or 2 mild or moderate events.

The dosage in our study (100/50 mg daily) is a commonly attainable dose in clinical practice. Zepatier has shown to be safe for subjects with chronic kidney disease or who are on hemodialysis. Less than 1% of Zepatier is excreted renally. In Merck C-SURFER, a phase 1 randomized, controlled Zepatier trial, subjects with advanced kidney disease tolerated the drug well for the required 12 weeks and had no need for dose adjustments.<sup>10</sup>

Zepatier trials have demonstrated a 94-100% success rate achieving HCV RNA levels of <15 IU/ml after 12 weeks of treatment (SVR-12) among genotype 1 or 4 HCV patients.<sup>3,4</sup>

HCV genotype (either on donor sera or recipient sera) will be confirmed by the standard of care diagnostic test at the Hospital of the University of Pennsylvania.

# 4.4. Mavryet or Epclusa for recipients of kidney transplants from donors with HCV infection that is genotype 2, 3, 5, or 6

For recipients transplanted with a kidney from a donor with genotype 2, 3, 5, or 6, the treatment regimen will be either 8 weeks of Mavyret (glecaprevir 100 mg and pibrentasvir 40 mg) or Epclusa (sofosbuvir 400 mg and velpatasvir 100 mg).

Mayvret is similar to Zepatier and has demonstrated SVR-12 (cure) rates of genotype 1 and 4 HCV of 99%.<sup>11</sup> Mavyret has additionally been shown to have cure rates of 95-99% in patients with genotypes 2, 3, 5, or 6, and thus is considered a pan-genotypic regimen.<sup>12</sup> Mavyret has been used to treat HCV in a broad range of populations including patients with chronic kidney disease and solid organ transplant recipients. Similar to

Zepatier, Mavyret has a favorable side effect profile and is safe to administer in the setting of renal dysfunction.<sup>13</sup> Mavyret is contraindicated with specific statin medications, including simvastatin and atorvastatin, for which reason Mavyret will not be used in patients taking these drugs. Mavyret may be inconsistently absorbed when crushed and administered via a feeding tube, for which reason the drug will only be started in the setting of a post-transplant patient who is extubated, stable, and taking medications.

The Epclusa treatment regimen, similar to Zepatier, has demonstrated SVR-12 (cure) rates of genotype 1 and 4 HCV that exceeds 95%. However, Epclusa has also been shown to have cure rates of 95-100% in patients with genotypes 2, 3, 5, or 6, and is thus considered a pan-genotypic HCV regimen. Epclusa has been shown to be safe to be administered in patients with renal dysfunction.

In the unlikely event that the patient has a contraindication to Mavyret and Epclusa, the investigators will identify and administer the safest and most effective alternative antiviral treatment.

In the unlikely event that neither the donor nor the recipient HCV can be genotyped, the investigators will identify and administer the safest and most effective pan genotypic regimen of either Mavyret or Epclusa.

### 5 CHAPTER 2: OBJECTIVES AND SPECIFIC AIMS

#### 5.1. Objectives

This study is being conducted to determine safety and efficacy of transplanting kidneys from HCV-NAT-positive donors into HCV-negative patients on the kidney transplant waitlist, who will then be treated with Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment post-transplantation.

#### 5.2. Specific aims

#### Primary aim:

- 1. <u>Primary efficacy objective</u>: to determine sustained virologic response (SVR) rates of open-label Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment in hepatitis C virus (HCV) negative patients who receive a kidney transplant from an HCV-infected donor, leading to post-transplantation de-novo HCV infection.
- 2. <u>Primary safety objective</u>: to determine the safety of administration of open-label Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment among HCV-negative patients who receive a kidney transplant from an HCV-infected donor and develop post-transplant HCV infection.

#### Secondary aims:

- 3. To determine 1-year graft survival rates of HCV-negative kidney transplant patients who receive a kidney transplant from an HCV-positive donor, including those who spontaneously clear HCV and those who receive open-label Zepatier, Mavyret, Epclusa, or another appropriate antiviral treatment upon development of de-novo HCV.
- 4. To evaluate rates of spontaneous clearance of HCV among HCV-negative patients who receive a kidney transplant from an HCV-infected donor.

### 6 CHAPTER 3: SCREENING AND SUBJECT SELECTION

#### 6.1. Recruitment: identification and screening process

The trial's phases can be categorized as "screening phase," (when patients are consented and will undergo evaluation for enrollment), "waiting list phase" (when patients are enrolled and are waiting for an offer of transplantation) and "transplantation phase" (after a HCV-positive kidney has been received and transplanted).

Subjects will be recruited for this pilot open-label clinical trial. Potential subjects will first be identified by the transplant nephrologist, clinical staff, and/or research staff evaluating patients at the transplant nephrology clinic at the University of Pennsylvania. There will be two key methods to identifying potential subjects. On the day of a patient's evaluation for waitlisting for a kidney transplant, the transplant nephrologist will identify patients as potential subjects for the study. Additionally, the research coordinator will review the kidney transplant waitlist every two weeks with a study investigator to identify potential subjects who have ≤2555 (blood group A, B, or O) and ≤1825 (blood group AB) days of waitlist or dialysis time by enrollment. Updates on transplant status will be continued to followed for these patients even after initial review and noted as apart of study data.

Potential subjects will be contacted via telephone by the research coordinator and/or research staff to gauge interest. In addition, we will obtain permission from the transplant nephrologists for their patient's participation, through hospital email. The nephrologists will be instructed in the e-mail that if we do not hear an objection within 48 hours, then that is commensurate to their assenting that their patient is appropriate for study participation. Potential subjects meeting inclusion and exclusion criteria will be invited to attend an informational meeting/presentation either in-person or by video conference (in accordance with University of Pennsylvania Office of Clinical Research regulatory guidance), where the study investigators and research staff will explain the study and its risks and benefits. If the patient is interested in participating in the study, informed consent will be acquired by the research staff, at which time the subject can formally be screened for entry.

Patients who are screened will be tracked in a pre-screening log to facilitate the screening process. The study team has worked with their department's Information Technology Team and their recommendations for protecting potential subject health information will be put into place.

During screening, the investigators will review the list of patient's medications and identify medications that might be contraindicated with potential direct acting antiviral treatments (example: atorvastatin, which interacts with Mavyret). If clinically appropriate, the investigators may recommend to the patient and primary provider to stop or change the medication in anticipation of future treatment for hepatitis C virus infection.

#### 6.1.1. Disenrollment criteria

Subjects who are designated status 7 (temporarily inactive and unable to receive any kidney offers until reactivated) will continue to be followed. If the subject is reactivated, his/her status, based on the inclusion and exclusion criteria, will be reviewed by the investigator team to ensure the patient is still eligible for the study. Additionally, as stated below, an inclusion criterion is ≤2555 days of accrued waiting time at the time of enrollment for blood group A, B, or O and ≤1825 days for blood group AB. If a subject remains enrolled at the time he/she has accrued 2920 days (for blood group A, B, or O) or 2190 days (for blood group AB) of waiting/priority time, he/she will be disenrolled, but will stay on the kidney transplant waiting list at Penn. If a subject reaches 66 years of age, he/she will be disenrolled from the study. Once a subject is disenrolled from the study, his/her UNOS status will be changed to reflect that they are no longer accepting hepatitis C-positive kidneys.

#### 6.2. Subject selection criteria

#### 6.2.1. Inclusion criteria

- Must be waitlisted for a kidney transplant (dialysis is not a requirement if a patient is waitlisted)
- Listed for an isolated kidney transplant with ≤2555 days of accrued transplant waiting time and/or
   ≤2555 days of dialysis time for blood group A, B, or O, by enrollment
- Listed for an isolated kidney transplant with ≤1825 days of accrued transplant waiting time and/or
   ≤1825 days of dialysis time for blood group AB, by enrollment
- No available living kidney donor
- Between 30-70 years of age
- Have a panel reactive antibody level ≤97%
- eGFR <15ml/min/1.73m<sup>2</sup> as calculated using the 4 variable MDRD equation
- Obtained agreement for participation from the patient's treating transplant nephrologist
- Able to travel to the University of Pennsylvania for routine post-transplant visits and study visits for a minimum of 6 months after transplantation
- No active illicit substance abuse
- Weigh at least 50kg
- Women must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) following transplant due to the increased risk of birth defects and/or miscarriage
- Both men and women must agree to use at least one barrier method to prevent any secretion exchange
- Inclusion criteria for treatment (not for entry as study patient) will include any detectable HCV RNA
- Able to provide informed consent

#### 6.2.2. Exclusion criteria

- Hepatocellular carcinoma
- Patients with primary focal segmental glomerulosclerosis (FSGS), FSGS recurring after previous transplant, or disease process with increased risk of causing early graft failure as per the treating nephrologist
- HIV positive
- HCV RNA positive (can be isolated HCV antibody positive provided the subject has no history of previously treated HCV)
- Hepatitis B surface antigen positive
- Any other chronic liver disease (excluding non-alcoholic fatty liver disease (NAFLD) with abnormal liver enzymes
- Persistently elevated liver transaminases
- Significant hepatic fibrosis on screening elastography (≥f2 fibrosis)
- Pregnant or nursing (lactating) women
- Known allergy or intolerance to tacrolimus that would require post-transplant administration of cyclosporine, rather than tacrolimus given the drug-drug interaction between cyclosporine and certain DAAs
- Waitlisted for a multi-organ transplant (e.g., pancreas-kidney, heart-kidney, etc.)

- Significant cardiomyopathy defined as either:
  - Left ventricular ejection fraction <40% on most recent echocardiogram</li>
  - Left ventricular ejection fraction ≥40% but <50% on most recent echocardiogram with an <5 METS of exercise tolerance</li>
  - Reversible ischemia on stress testing without revascularization

#### 6.3. Donor Organ Selection Criteria

#### **Inclusion Criteria**

- Detectable HCV RNA
- Age ≤60 years
- Study *modified* Kidney donor profile index (KDPI) score ≤0.85<sup>6</sup> calculated as if the kidney were HCV-negative (https://optn.transplant.hrsa.gov/resources/allocation-calculators/kdpi-calculator/)

#### **Exclusion Criteria**

- Anatomical issues in the kidney allograft that raise the risk of post-transplant complications (e.g., number or length of renal arteries or veins)
- Confirmed HIV positive
- Confirmed HBV positive (positive Hepatitis B surface antigen and/or HBV DNA)
- Known previously failed treatment for HCV using a regimen with a direct-acting antiviral (can have received interferon monotherapy and/or interferon + ribavirin combination therapy)

#### 6.3.1. Donor Evaluation

To remain in the study, subjects will receive a kidney transplant from a confirmed HCV-infected donor as demonstrated by HCV NAT results reported by UNOS or the organ procurement organization.

#### 6.3.2. Donor Genotyping (when possible)

We will accept donor or recipient HCV genotype results for guidance of appropriate antiviral therapy for recipients. The ability to obtain donor blood for HCV genotype testing prior to transplant will not be required.

Where available, donor genotyping will be performed on specimens provided to the Molecular Pathology Laboratory by LABS and Gift-of-Life, the local organ procurement organization. These specimens will be taken from potential kidney donors once the organ procurement organization has been notified of the potential donor and will be qualified for testing by Gift-of-Life.

In other instances, we will perform genotyping of the kidney recipient in the first week after transplantation. The assay that will be used for HCV genotyping is a laboratory-developed assay that was validated by the HUP MPL under the guidance of Vivianna Van Deerlin, MD, PhD. The validation process entailed testing multiple past clinical samples with known HCV genotypes, as well as purchased HCV genotype controls, and assessing concordance between the results obtained and the expected results. <sup>16</sup> This assay (the eSensor® HCVg *Direct* Test, GenMark Diagnostics) has also been validated by multiple external laboratories with the following results: Covance Central Laboratory Services (482 samples, 98.6% concordance), University of Minnesota (135 samples, 96.4% concordance), and the University of Washington (77 samples, 97.4%). <sup>17-19</sup> In the HUP MPL, overall, the assay was able to genotype all purchased controls correctly (n=15, HCV genotypes 1 through 6, concordance = 100%). It was also able to correctly genotype the vast majority of prior clinical samples (n=56 of 61, HCV genotypes 1 through 6, concordance = 92%). Resolution of discordant samples showed that the limitations of the assay, as determined by the validation, included decreased ability to genotype samples with: low viral loads, mixed genotype infections, or HCV genotype 4f infection. These limitations are felt to be minor as low viral loads

specimens are not expected from HCV-untreated organ donors, and mixed genotype / genotype 4f specimens are very rarely encountered in the United States. The validation samples were picked to better understand the limitations of the assay and so had a higher proportion of mixed infection samples (n=6) and rare genotype samples (e.g., Type 4f, n=1) than what is encountered clinically. A retrospective review by the MPL of HCV genotypes resulted at HUP over a 14-month period (July 2014 to October 2015) by the previous MPL HCV genotyping assay (Siemens VERSANT HCV Genotype 2.0) found a total of 6 mixed infections and one genotype 4f infection out of 1,551 samples tested (~0.4% and 0.06%, respectively).

#### 6.3.2. Drug Resistance Testing

Participants with Genotype 1a and Genotype 1 HCV infection with an unknown subtype will have baseline NS5A drug resistance assay testing checked at the start of treatment. The Hepatitis C Viral RNA Genotype 1 NS5a Drug Resistance test will be used to check for NS5A drug resistance. This test uses reverse transcription polymerase chain reaction (PCR) and DNA sequencing to detect mutations [resistance associated variants (RAVs)] in the NS5a inhibitors. It has not been cleared or approved by FDA but has been validated pursuant to the CLIA regulations. The test will be performed by a lab qualified by the Principal Investigator Team. It has an analytical sensitivity of >95% for viral loads ≥1800 IU/mL.<sup>20</sup> Reported results include mutations and polymorphisms associated with NS5A inhibitor resistance (only if HCV genotype 1a, 1b, or 1 detected) as well as a patient specific interpretation:

- Resistance predicted: ≥1 mutation predicting NS5A inhibitor resistance detected
- Resistance not predicted: no mutations predicting NS5A inhibitor resistance detected

### 7 CHAPTER 4: TREATMENTS

#### 7.1. Zepatier (grazoprevir and elbasvir) for kidney recipients with HCV genotype 1 or genotype 4 infection

Zepatier tablets will be provided by Merck as part of this investigator-initiated protocol funded by Merck. Open-label Zepatier (grazoprevir 100 mg and elbasvir 50 mg) will be administered once daily by mouth for 12 weeks. An exception to the 12 week course of treatment will be if patients have polymorphisms at positions M28, Q30, L31, and/or Y93 as determined by the Hepatitis C Viral RNA Genotype 1 NS5a Drug Resistance test. In this case, treatment with Zepatier will be extended to 16 weeks and renally-adjusted Ribavirin will be initiated at the clinician's discretion, and continued for the remainder of therapy (until the 16-week mark). Such a strategy will provide optimal treatment, without delaying therapy prior to receipt of results of NS5A drug resistant testing. Grazoprevir (GZR)/ elbasvir (EBR) is a fixed-dose combination tablet without ribavirin.

GZR is an HCV ns3/4a inhibitor while EBR is an HCV NS5A inhibitor. Both are direct-acting antivirals, which together form an effective therapy for HCV virus and reduce the likelihood and effects of long-term liver-related HCV complications. GZR/EBR exhibits broad in vitro activity against most HCV genotypes and in vitro activity against many clinically relevant resistance-associated variants (RAVs).

Zepatier (GZR/EBR) has been evaluated globally in multiple phase I, II, and III trials to treat HCV. Randomized, placebo-controlled trials have been completed and led to obtain FDA approval for Zepatier as a treatment for genotype 1 or 4 HCV. As of July 1, 2015, a diverse population of over 1000 HCV patients has been exposed to Zepatier either as a single agent or in combination with ribavirin or sofosbuvir in phase I/II/III studies. Zepatier has been generally well tolerated at doses of 50-100 mg GZR and 50 mg EBR orally once daily. It has been comparably effective across all subgroups it has been tested in, including non-cirrhotic and/or treatment-naïve subjects.

Headaches, fatigue, and nausea represent the most common adverse drug reactions with Zepatier. Other drug-related adverse events have included arthralgia, insomnia, diarrhea, dizziness, pyrexia, and asthenia. Drug-related serious adverse events are uncommon, but include allergic reactions, possible adverse interactions with other medications, or elevated liver enzymes. In past Zepatier trials, the majority of the adverse events were reversible. These adverse events are usually grade 1 or 2 mild or moderate events.

The dosage in our study (100/50 mg qd) is a commonly attainable dose in clinical practice. Zepatier has shown to be safe for subjects with chronic kidney disease or who are on hemodialysis. Less than 1% of Zepatier is excreted renally. In Merck C-SURFER, a phase 1 randomized, controlled Zepatier trial, subjects with advanced kidney disease tolerated the drug well for the required 12 weeks and had no need for dose adjustments.

Zepatier trials have demonstrated a 94-100% success rate achieving HCV RNA levels of <15 IU/ml after 12 weeks of treatment (SVR-12) among genotype 1 or 4 HCV patients.

As of January 2016, Zepatier was approved by the Food and Drug Administration. It has been extensively studies in multiple large clinical trials. This drug regimen was chosen as first-line therapy, rather than other approved agents (i.e., Sofosbuvir/Ledipasvir, trade name Harvoni), as Zepatier has been shown to be safe and efficacious in patient with significant renal dysfunction. As a result, if a subject's kidney function has not fully recovered when treatment is initiated, the investigational agents can safely be administered, unlike other approved agents.

#### 7.?. Mavyret for kidney recipients with HCV genotypes 2, 3, 5, or 6 infection

For recipients transplanted with a kidney from a donor with genotype 2, 3, 5, or 6, we will consider a treatment regimen of 12 weeks of Mavyret (glecaprevir 100 mg and pibrentasvir 40 mg). This would be administered as 3 pills taken once daily for 8 weeks.

Glecaprevir (G) is a NS3/4A protease inhibitor, while pibrentasvir (P) is a NS5A inhibitor. Both are direct acting antivirals that have a high barrier to resistance in vitro and in combination have synergistic antiviral activity. G/P has been evaluated globally in multiple phase I, II, and III trials and has been approved by the FDA to treat all six HCV genotypes. It has been studied as a single agent and in combination with ribavirin. It has been effective across all sub-types, including treatment experienced and patients with cirrhosis.

The dosage in our study (3 pills of 100/40 mg qd) is a commonly attainable dose in clinical practice. Mavyret has shown to be safe for subjects with chronic kidney disease or who are on hemodialysis without any need to dose adjust. Mavyret is primarily cleared by the biliary system and a negligible amount is cleared by the kidneys. In EXPEDITION-4, a phase 3 multicenter open-label trial, subjects with advanced kidney disease tolerated Mavyret well for the required 8 weeks and had no need for dose adjustments and the drug was shown the have excellent efficacy with SVR rates of > 98%.

The most common side effects documented with Mavyret were headaches, fatigue, and less commonly nausea. Drug-related serious adverse events are uncommon, but include allergic reactions, possible adverse interactions with other medications, or elevated liver enzymes. In past Mavyret trials, the majority of the adverse events were reversible. These adverse events are usually grade 1 or 2 mild or moderate events.

Mavyret trials have demonstrated a 95-100% success rate achieving HCV RNA levels of <15 IU/ml after 12 weeks of treatment (SVR-12) among patients with HCV genotypes 1-6. It was approved for the treatment of hepatitis C genotypes 1-6 by the FDA in 2017.

A special consideration for Mavyret is that the drug's absorption may be impaired if crushed. For that reason, we will avoid administering the medication through a feeding tube. A second consideration is contraindicated medications including simvastatin and atorvastatin. These medications will not be co-administered with Mavyret.

### 7.?. Epclusa for kidney recipients with HCV genotypes 2, 3, 5 or 6 infection

For recipients transplanted with a kidney from a donor with genotype 2, 3, 5, or 6, we also will will consider a treatment regimen of 12 weeks of Epclusa (sofosbuvir 400 mg/velpatasvir 100 mg). This treatment regimen, similar to Zepatier, has demonstrated SVR-12 (cure) rates of genotype 1 and 4 HCV that exceeds 95%. However, Epclusa has also been shown to have cure rates of 95-100% in patients with genotypes 2, 3, 5, or 6, and is thus considered a pan-genotypic HCV regimen.

Sofosbuvir is an NS5B polymerase inhibitor and velpastasvir is a NS5A inhibitor. Both are direct acting antivirals that have a high barrier to resistance in vitro and in combination have synergistic antiviral activity. G/P has been evaluated globally in multiple phase I, II, and III trials and has been approved by the FDA to treat all 6 HCV genotypes. It has been studied as a single agent and in combination with ribavirin. It has been effective across all sub-types, including treatment experienced and patients with cirrhosis.

Epclusa has been shown to be safe to be administered in patients with renal dysfunction.<sup>21,22</sup> For individuals with renal impairment (GFR <30), we know that velpatasvir pharmacokinetics are not impacted. However, for inidivudals with a GFR <30 sofosbuvir can potentially accumulate and historically individuals with

17

CKD were excluded from trials. Sofosbuvir has been used off label in real-world case series without any safety concerns identified. A phase II single arm study of sofosbuvir/velpatasvir with 50 patients on hemodialysis showed that the drug was safe and well tolerated with SVR rates >95%.

Epclusa trials have demonstrated a 95-100% success rate achieving HCV RNA levels of <15 IU/ml after 12 weeks of treatment (SVR-12) among patients with HCV genotypes 1-6. Epclusa was approved by the FDA for treatment of hepatitis C genotypes 1, 2, 3, 4, 5, and 6 in 2016.

#### 7.1.1. Administration of Zepatier

Merck & Co will manufacture, package, and label Zepatier drug that will be provided to recipients with HCV genotype 1 and 4 infection. Each subject will receive a minimum of six bottles with each bottle containing a 14-day supply (14 capsules) of 100/50 mg Zepatier tablets. Daily dose will be one tablet.

The Investigational Drug Services (IDS) pharmacy, directed by Kenneth Rockwell, PharmD, will only be required to store and distribute the study drug. Sofosbuvir and Ribavirin will be purchased and sourced locally. Both of these medications will be purchased and stored by the IDS pharmacy at Penn. Ribavirin will be generic and the manufacturer will vary depending on monthly price fluctuations.

Zepatier will be picked up from the investigational drug services (IDS) pharmacy by the research staff at 28-day intervals. The study staff will deliver the medication to the subjects at their study visits (patients expected to be at home by the time that HCV therapy is initiated and patients will be given medication at their scheduled post-transplant/study visit). Treatment with the study drug will begin within 4 weeks post-transplant. If hepatitis C is not cured after a subject has received Zepatier, he or she will be treated with a second regimen that includes Zepatier plus Sovaldi (Sofosbuvir) and Ribavirin. Any patient (male or female) receiving ribavirin as part of the first- or second-line regimen will be required to use two methods of birth control while on Ribavirin therapy, with continuing two forms of birth control for up to 6 months after the last dose of the study drug.

#### 7.1.2. Drug logistics and accountability

Study medication bottles must be stored according to the medication label. Study drug must be protected from moisture. The research staff or investigator will instruct the subject on the proper administration of Zepatier. Zepatier tablets should be taken once daily by mouth. The investigator, or a responsible party designated by the investigator, must maintain a careful record of the inventory and disposition of the investigational agent using the drug accountability form. If a subject loses the bottle of study medication, the research staff should contact Kenneth Rockwell, Pharmacist at the research pharmacy. A replacement bottle with the appropriate amount of study medication will be made available at the research pharmacy.

#### 7.1.3. Destruction and return

At the conclusion of the study, remaining medication from the study patients (and left-over medication) will be destroyed at the clinical site, after approval is granted by the research pharmacy for the drug destruction plan. Destruction will be documented in the drug accountability form.

#### 7.1.4. Zepatier Initial Treatment Failures

Study subjects with treatment failure, defined as virologic breakthrough (when an undetectable viral load while on treatment becomes detectable or a ≥ one log increase from nadir HCV RNA) or virologic relapse (undetectable viral load after completion of treatment that during the 12-week post-treatment follow-up period becomes detectable) will be provided open-label Zepatier + Sofosbuvir (Sovaldi) 400 mg + Ribavirin (generic), renally dosed based on creatinine clearance per the manufacturer guidelines. Any subjects who experience treatment failure will repeat the original study lab visit and visit protocol once they begin their secondary

treatment with Zepatier, sofosbuvir, and ribavirin, similar to subjects initiating HCV treatment following kidney transplantation. Prior to initiating treatment with this regimen, patients will have serum NS5A resistance (RAV) testing.

#### 7.2. Administraton of Mavyret or Epclusa for kidney recipients with genotype 2, 3, 5, or 6 HCV infections

Upon receiving the results of genotype testing of the donor and/or kidney recipient showing HCV infection that is neither genotype 1 nor genotype 4 (genotypes 2, 3, 5 or 6), PIs will coordinate treatment with Mavyret or Epclusa that will be locally sourced by the hospital pharmacy. In the unlikely event that the patient has a contraindication to Mavyret or Epclusa, another optimal antiviral regimen will be selected.

The Hospital of the University of Pennsylvania (HUP) will provide the antiviral treatment and coordinate the application to the subject's insurance company for coverage of the antiviral treatment. In the event that the subject's insurance company denies coverage for the antiviral treatment, HUP will provide the entire HCV treatment regimen at no charge to the subject. In the event that the subject fails to be cured of HCV with the initial treatment regimen and the subject's insurance declines to pay for a second antiviral treatment, HUP will provide the second HCV treatment regimen at no charge to the subject.

### 8 CHAPTER 5: DATA COLLECTION

#### 8.1. Study visits

Study visits are scheduled to occur following subjects' standard post-transplant follow-up visits. Since treating nephrologists do not always require stable post-transplant patients to attend these visits, subjects may be asked to come in solely for study visits. These visits will be encouraged, but not required unless the study drug is being dispensed that day. For all other study visits, a missed visit by a stable subject who has had necessary labs drawn will not be considered a protocol violation.

#### 8.1.1. Informed consent

During the screening phase, potentially eligible, interested subjects will be invited to attend an informational session/presentation either in-person or by video conference, consistent with University guidelines. The following procedures will be performed during the screening process:

- Sign and date the ICF and HIPAA authorization this signing can be done in-person or electronically (eSign) using University approved procedures (e.g., REDCap)
- Review of inclusion/exclusion criteria
- Schedule for screening visit

After completing the informational session and signing the informed consent, the subject will be scheduled for a screening visit within 56 days if the subject meets inclusion/exclusion criteria thus far. The study staff will call the subject 1-2 days prior to the screening visit and send a reminder letter as well if the screening visit is not conducted within the 2 weeks following consent. The study staff will instruct the subject to not eat or drink (except water) and to avoid heavy exercise for 3 hours prior to the study visit in order to ensure accuracy of the Fibroscan test that requires 3 hours of NPO prior to testing. According to the recommendations of use and based on safety and efficacy matters; patients with ascites (fluid in the abdomen), persons with active implantable medical devices, and persons with a waist size more than 100cm will be excluded from having a Fibroscan performed.

#### 8.1.2. Screening

The following procedures and activities will be performed during the screening process, after the informed consent is signed:

- Review medical history
- Vital signs
- Physical exam
- Fibroscan
- Review current medications
- Labs/phlebotomy: hepatic function panel, HCV RNA, HBV DNA, and HIV antibody if these labs have not been checked within the last 365 days, as per the transplant center protocol for yearly testing of these labs (to ensure patients are up to date with the all center requirements for lab testing)
- Updated transthoracic echocardiogram if one is needed for a patient to remain updated as per the transplant center protocol
- Completion of health status questionnaire (RAND-36)
- Provide instructions on recording of new medications and dose changes

#### 8.1.3. Post-Kidney Transplant

#### 8.1.3.1. Post-Kidney Transplant Visits

Patients, after receiving a kidney transplant are followed very closely by both the surgical and nephrology team.

As apart of standard of care visits, the following procedures activities will be performed:

- Phlebotomy
- Vital signs
- Physical exam

The study staff will follow procedures and activities closely along with transplant team and this information (vital signs, physical exam, and phlebotomy results) will be collected as apart of data collection. In addition to these standard of care procedures and activities, the study team will also perform specific research related activities at specific time points.

#### 8.1.3.2. Post-Kidney Transplant Research Phlebotomy

Research laboratory blood draws will take place along with standard of care blood draws outlined in Section 8.2.1. The study staff will call the research subject to coordinate research blood draws appropriately. In addition, study staff will assess for adverse events/side effects and obtain current medication data.

As outlined in Section 8.2.1, patients with a positive HBV Core Antibody, HBV-DNA levels will be checked every 6 weeks while on Zepatier and LFTs will be closely monitored. HBV therapy may be considered the transplant team as medically appropriate.

Additional laboratory testing will be done if the PIs feel it is necessary for patient safety.

#### 8.1.3.3. Visit 1: Post-kidney transplant (between days 2 – 7)

The study staff will meet the subject in their HUP hospital room, three days after their kidney transplant.

#### Initiating antiviral treatment

Treatment with the study drug will begin when the patient has a detectable HCV RNA post-transplantation and the donor and/or recipient have had an HCV genotype ascertained to guide treatment. As appropriate, subjects being discharged will be provided with a sufficient supply of the study drug and instructed to begin treatment once HCV RNA is confirmed, which may occur any time between weeks 1-4. When the subject begins treatment for HCV, the staff will notify the subject's primary nephrologist and primary care physician. During the initial hospitalization, the HUP pharmacy staff will commence the process of assessing the patient's insurance and first-line DAA regimen in the event of an HCV genotype that is not appropriate for Zepatier treatment.

As with any scientific protocol, safety will be considered before treating the patients. The treating physician will evaluate the patient's overall condition and make a judgment on whether initiating treatment is safe.

The following research procedures and activities will be performed:

- Assess for Adverse Events
- Obtain medication data
- Research Phlebotomy, including the NS5A drug resistance assay testing as appropriate (See Section 8.2.1 for complete list)

Dispense study drugs

Blood samples for immunologic t-cell assays will be processed and banked or shipped.

#### 8.1.3.3.1. Management of patients with genotype 1 HCV and NS5A resistance variants

Once HCV infection is confirmed, patients will have their HCV genotype reconfirmed. Patients with Genotype 1a and Genotype 1 with an unknown subtype will have baseline NS5A drug resistance assay testing. This will be checked at start of treatment. If patients have polymorphisms at positions M28, Q30, L31, and/or Y93, treatment with Zepatier will be extended to 16 weeks, rather than 12 weeks, and renally-adjusted Ribavirin at the clinician's discretion will be initiated, and continued for the remainder of therapy (until the 16 week mark). Such a strategy will provide optimal treatment, without delaying therapy prior to receipt of results of NS5A drug resistant testing. Under such a scenario, all of the study procedures referenced above and below will be extended by 4 weeks. Any patient (male or female) receiving ribavirin as part of the first- or second-line regimen will be required to use two methods of birth control while on Ribavirin therapy, with continuing two forms of birth control for up to 6 months after the last dose of the study drug.

#### 8.1.3.4. Visit 2: (day $10 \pm 2$ day)

Visit #2 should occur  $10 \pm 1$  days after the subject's kidney transplant and will immediately follow the subject's regularly scheduled post-transplant follow-up visit. The staff will call the subject 1-2 days before the visit. During this phone call, the research staff will remind the subject where to go for the study visit, to take their routine and study medications as they usually would prior to the visits and if a Fibroscan is needed, inform the subject and remind him/her to not eat or drink for three hours before the study visit.

The subject will arrive at the study site outpatient clinic. The following procedures and activities will be performed:

- Assess for Adverse Events
- Obtain medication data
- Research Phlebotomy (See Section 8.2.1 for complete list)
- Pill count and verbal assessment for drug adherence
- Schedule appointments for follow-up visits

The study staff will reinforce instructions on bringing the subject's routine and study medications to each visit, will thank the subject for their attendance, and reinforce adherence with the study medication and protocol.

#### 8.1.3.5. Visit 3: (day $21 \pm 3$ days)

Visit #3 should occur three weeks ( $21\pm3$  days) after the subject's kidney transplant and will immediately follow the subject's regularly scheduled post-transplant follow-up visit. The staff will call the subject 1-2 days before the visit. During this phone call, the research staff will remind the subject where to go for the study visit, to take their routine and study medications as they usually would prior to the visits and if a Fibroscan is needed, inform the subject and remind him/her to not eat or drink for three hours before the study visit.

The subject will arrive at the study site outpatient clinic. The following procedures and activities will be performed:

- Assess for Adverse Events
- Obtain medication data

- Research Phlebotomy (See Section 8.2.1 for complete list)
- Pill count and verbal assessment for drug adherence
- Schedule appointments for follow-up visits

#### 8.1.3.6. Visit 4 (day $28 \pm 3$ days)

Visit #4 should occur 4 weeks ( $28 \pm 3$  days) after the subject's kidney transplant and will immediately follow the subject's regularly scheduled post-transplant follow-up visit. The staff will call the subject 1-2 days before the visit. During this phone call, the research staff will remind the subject where to go for the study visit, to take their routine and study medications as they usually would prior to the visits and if a Fibroscan is needed, inform the subject and remind him/her to not eat or drink for three hours before the study visit.

The subject will arrive at the study site outpatient clinic. The following procedures and activities will be performed:

- Assess for Adverse Events
- Obtain medication data
- Research Phlebotomy (See Section 8.2.1 for complete list)
- Fibroscan (elastography of liver)
- Completion of health status questionnaire (RAND-36) (to assess changes in health status from preto post-transplant)
- Pill count and verbal assessment for drug adherence
- Replenish study drug as appropriate with the DAA prescribed from the specialty pharmacy

#### **HCV Non-Transmission**

It is possible that a subject may not develop chronic HCV infection, either due to non-transmission or spontaneous clearance of HCV by week 4 (defined as an initial positive HCV RNA and subsequent undetectable HCV RNA without treatment). If a subject has an undetectable HCV RNA based on the week 4 HCV RNA, a repeat HCV RNA will be checked at week 8 to ensure non-infection with HCV, rather than a false-negative HCV RNA. If the week 8 HCV RNA confirms lack of infection (undetectable week 8 HCV RNA), then no further treatment will be needed. Subjects will be assessed at a study visit and HCV RNA levels re-checked at week 16 and 28 post-kidney transplantation. Should any subject spontaneously clear HCV without treatment, another subject will replace them in order to meet our planned treatment sample size of 10.

#### 8.1.3.7. Visits 5 & 6 (day 42±7, day 56±7)

Visit #5 should occur 6 weeks (42±7 days) after the subject's kidney transplant and will immediately follow the subject's regularly scheduled post-transplant follow-up visit. Visit #6 should occur 8 weeks (56±7 days) after the subject's kidney transplant and will immediately follow the subject's regularly scheduled post-transplant follow-up visit.

For both visits, the staff will call the subject 1-2 days before the visit to remind subject of visit. During this phone call, the research staff will remind the subject where to go for the study visit, to take their routine and study medications as they usually would prior to the visits and, if a Fibroscan is needed, inform the subject and remind him/her to not eat or drink for three hours before the study visit.

The following procedures and activities will be performed:

- Assess for Adverse Events
- Obtain medication data
- Research Phlebotomy (See Section 8.2.1 for complete list)

- Replenish study drug
- Pill count and verbal assessment for drug adherence

As needed, the staff will replenish the subject's supply of the DAA sometime during visits #4 & 5, depending on when the subject began treatment. For Mavyret, the treatment course is expected to be 8 weeks.

#### 8.1.3.8. Visits 7 & 8 (day 87 + 7, day 112 + 14)

Visit #7 should occur 12 weeks (87 + 7 days) after the subject's kidney transplant and will immediately follow the subject's regularly scheduled post-transplant follow-up visit. Visit #8 should occur 16 weeks (112 + 14 days) after the subject's kidney transplant and will immediately follow the subject's regularly scheduled post-transplant follow-up visit.

Midway between these study visits, subjects will be phoned in order to ensure drug adherence, if necessary

For both visits, the staff will call the subject 1-2 days before the visit to remind subject of visit. During this phone call, the research staff will remind the subject where to go for the study visit, to take their routine and study medications as they usually would prior to the visits and, if a Fibroscan is needed, inform the subject and remind him/her to not eat or drink for three hours before the study visit.

The following procedures and activities will be performed:

- Assess for Adverse Events
- Obtain medication data
- Research Phlebotomy (See Section 8.2.1 for complete list)
  - Note: Timing for HCV RNA viral load, post treatment, should, as best possible, follow the important data collection points post treatment. These are as follows:
    - Post-treatment: This should occur after the subject has completed treatment of the study drug.
    - SVR 4: This should occur 4 weeks after the subject has completed treatment.
    - SVR 8: This should occur 8 weeks after the subject has completed treatment.
    - SVR 12: This should occur 12 weeks after the subject has completed treatment.
    - SVR 24: This should occur 24 weeks after the subject has completed treatment.
- Fibroscan (elastography of liver) for Visit 8 only
- Completion of health status questionnaire (RAND-36) (to assess changes in health status from preto post-transplant)
- Pill count and verbal assessment for drug adherence
- Replenish study drug
  - Note: The staff will replenish the subject's supply of the DAA between visits 7 & 8, if necessary. This is based on management of patients NS5A resistance variants, in any were/are present. The staff will also remind the subject how to take the medication, for those subjects still on study medication.

#### 8.1.3.9. Visit 9 (day 140 ±7)

Visit #9 should occur 12 weeks (140  $\pm$ 7 days) after the subject's kidney transplant and will immediately follow the subject's regularly scheduled post-transplant follow-up visit.

For this visit, the staff will call the subject 1-2 days before the visit. During this phone call, the research staff will remind the subject where to go for the study visit, to take their routine and study medications as they usually would prior to the visits and if a Fibroscan is needed, inform the subject and remind him/her to not eat or drink for three hours before the study visit.

The following procedures and activities must be performed:

- Assess for Adverse Events
- Research Phlebotomy (See Section 8.2.1 for complete list)
  - Note: Timing for HCV RNA viral load, post treatment, should, as best possible, follow the important data collection points post treatment. These are as follows:
    - Post-treatment: This should occur after the subject has completed treatment of the study drug.
    - SVR 4: This should occur 4 weeks after the subject has completed treatment.
    - SVR 8: This should occur 8 weeks after the subject has completed treatment.
    - SVR 12: This should occur 12 weeks after the subject has completed treatment.
    - SVR 24: This should occur 24 weeks after the subject has completed treatment.
- Fibroscan (elastography of liver)
- Complete a health status questionnaire (RAND-36)

#### 8.1.3.10. Visit 10 (day 365 ±14)

Visit #10 should occur 52 weeks (365 ±14 days) after the subject's kidney transplant and will immediately follow the subject's regularly scheduled post-transplant follow-up visit.

For this visit, the staff will call the subject 1-2 days before the visit. During this phone call, the research staff will remind the subject where to go for the study visit, to take their routine and study medications as they usually would prior to the visits and, if a Fibroscan is needed, inform the subject and remind him/her to not eat or drink for three hours before the study visit.

The following procedures and activities must be performed:

- Assess for Adverse Events
- Research Phlebotomy (See Section 8.2.1 for complete list)
- Fibroscan (elastography of liver)
- Complete a health status questionnaire (RAND-36)

The Research Staff should fill out the **Study Closeout Form.** This form must be signed by the principal investigator.

#### 8.1.3.11. Additional Visits

Additional visits will only be necessary in the case of treatment failures. If treatment failure occurs, subjects with genotype 1 or 4 infections will be treated with Zepatier and two other hepatitis C medications, Sofosbuvir (Sovaldi), and Ribavirin for an additional 12 weeks. All study and lab visits will be repeated during this secondary treatment period. NS5A resistance (RAV) testing will be checked again (a second time) prior to initiating second-line therapy.

If treatment failure occurs for patients with non-genotype 1 and non-genotype 4 infections (i.e. genotypes 2, 3, 5, or 6), the PIs will evaluate these patients for second treatment regimen that will be paid for either by the patient's insurance company or provided by HUP if the insurance company denies payment.

#### 8.1.5. Long-term outcomes and Future research

We will collect long-term outcome data beyond the end of the 12-month active study participation period. We will passively monitor care through the electronic medical record in order to identify and track problems with organ function or other health problems that may develop, related to the transplant and study participation. This data will be stored safely like all other data, with all necessary precautions.

Subjects will also be approached to provide optional blood sample for testing of viral kinetics (HCV RNA), donor and recipient IL-28B polymorphisms, and alloimmune responses (T- and B-cell function). Samples will be stored in a locked freezer, using encrypted patient IDs.

De-identified samples from subjects may be sent to other investigators for their research. These samples may include information such as sex, age, health history, or ethnicity. These samples will not be sold. Some future studies may need health information (such as smoking history or present health status) that may require contacting the subject to obtain.

### 8.2. Study schedule of procedures

### 8.2.1. Visits, lab testing, and other clinical testing

| THINKER Summary of | f Study Activities | – Zepat | ier or I | Epclus | а | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Visit | Sched | ule | | Res | earch | Visit / | Activities | Research Labs | | | | | | | Standard of Care | | | |
| Week(s) post-KT | Day(s) post-<br>KT | Visit | Study Visits | Fab-Only | Informed Consent | Assess Adverse Events | Current Medications | Fibroscan | RAND-36<br>Health Status<br>Questionnaire | HBV SA, HIV AB, & LFTs | HBV Core Antibody | Urine Preg Test | HCV RNA | Viral Kinetics (optional)◆ | NS5A Resistance** | Genotyping of donor<br>and/or recipient | Vitals &<br>Physical Exam | *dMD | эвэ | Tacrolimus |
| Screening | | | | | / | 1 | 1 | / | ✓ | ✓ | ✓ | 1 | 1 | | | | ✓ | | | |
| 1 (Begin treatment) | Day 2 - 7 | V1 | 1 | | | 1 | 1 | | | | ✓• | | 1 | 1 | 1 | 1 | ✓ | ✓ | ✓ | 1 |
| 1 | 7 ± 1 day | | | ✓ | | | 1 | | | | | | 1 | 1 | | | | ✓ | ✓ | 1 |
| 2 | 10 ± 1 day | V2 | ✓ | | | 1 | ✓ | | | | | | 1 | 1 | | | ✓ | ✓ | ✓ | 1 |
| 2 | 14 ± 1 day | | | ✓ | | | ✓ | | | | | | 1 | 1 | | | | ✓ | ✓ | ✓ |
| 3 | 21 ± 3 day | V3 | ✓ | | | 1 | ✓ | | | | | | ✓ | 1 | | | ✓ | 1 | 1 | ✓ |
| 4 | 28 ± 3 day | V4 | ✓ | | | 1 | ✓ | ✓ | ✓ | | | | ✓ | ✓ | | | ✓ | 1 | 1 | ✓ |
| 6 | 42 ± 7 day | V5 | 1 | | | 1 | 1 | | | | ✓• | | 1 | 1 | | | ✓ | <b>✓</b> | <b>✓</b> | <b>\</b> |
| 8 | 56 ± 7 day | V6 | 1 | | | 1 | 1 | | | | | | 1 | 1 | | | 1 | 1 | 1 | 1 |
| 10 | 70 ± 3 day | | | 1 | | 1 | 1 | | | | | | | 1 | | | | 1 | 1 | 1 |
| 12 | 84 ± 14 day | V7 | 1 | | | 1 | 1 | | | | ✓• | | | 1 | | | 1 | 1 | 1 | 1 |
| 13<br>(End treatment)† | 87 + 7 day | | | 1 | | | 1 | | | | | | 1 | 1 | | | | | | |
| 16† (SVR 4) | 115 + 14 day | V8 | 1 | | | 1 | 1 | | ✓ | | | | 1 | 1 | | | 1 | 1 | 1 | 1 |
| 20 (SVR 8) | 140 ±7 day | | | 1 | | | | | | | | | 1 | 1 | | | | ✓ | ✓ | 1 |
| 24 (SVR 12) | 171 +14 day | V9 | 1 | | | 1 | | 1 | ✓ | | | | 1 | 1 | | | 1 | 1 | 1 | 1 |
| 28 | 196 ±7 day | | | 1 | | | | | | | | | | 1 | | | | 1 | 1 | 1 |
| 32 | 224 ±7 day | | | 1 | | | | | | | | | | 1 | | | | 1 | 1 | 1 |
| 36 (SVR 24) | 252 ±7 day | | | 1 | | | | | | | | | 1 | 1 | | | | 1 | 1 | 1 |
| 40 | 280 ±14 day | | | 1 | | | | | | | | | | 1 | | | | 1 | 1 | 1 |
| 52 | 365 ±14 day | V10 | 1 | | | 1 | | 1 | / | | | | 1 | 1 | | | 1 | 1 | 1 | 1 |

<sup>\*</sup> CMP=comprehensive metabolic panel which includes basic metabolic panel and liver function tests \*\*As needed \$\display\text{Viral Kinetics testing can be done anytime there is a standard of care blood draw \$\display\text{If patients require the 16 weeks of therapy, the last 4 weeks would be the same as weeks 9-12 of therapy. If patients require only 8 weeks of therapy, then the lab test schedule will be modified to calculate SVR 4, 8 and 12 based on end of therapy

Only if HBV Core Antibodies are positive.

| THINKER Summary of | f Study Activities | – Mavv | ret | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 7 7 10 11 11 10 | | Sched | ule | | Res | earch | Visit A | Activities | | Research Labs | | | | | | Standard of Care | | | |
| Week(s) post-KT | Day(s) post-<br>KT | Visit | Study Visits | Lab-Only | Informed Consent | Assess Adverse Events | Current Medications | Fibroscan | RAND-36<br>Health Status<br>Questionnaire | HBV SA, HIV AB, & LFTs | HBV Core Antibody | Urine Preg Test | HCV RNA | Viral Kinetics (optional)◆ | NS5A Resistance** | Genotyping of donor<br>and/or recipient | Vitals &<br>Physical Exam | CMP* | СВС | Tacrolimus |
| Screening | | | | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | 1 | ✓ | | | | <b>√</b> | | | |
| 1 (Begin treatment) | Day 2 - 7 | V1 | 1 | | | 1 | 1 | | | | ✓• | | 1 | 1 | 1 | ✓ | ✓ | 1 | 1 | 1 |
| Treatment Week 1 | 7 ± 1 day | | | 1 | | | 1 | | | | | | 1 | 1 | | | | 1 | 1 | 1 |
| Treatment Week 2 | 10 ± 1 day | V2 | 1 | | | 1 | 1 | | | | | | 1 | 1 | | | ✓ | 1 | 1 | 1 |
| 2 | 14 ± 1 day | | | 1 | | | 1 | | | | | | 1 | 1 | | | | 1 | 1 | 1 |
| Treatment Week 3 | 21 ± 3 day | V3 | 1 | | | 1 | 1 | | | | | | 1 | 1 | | | ✓ | 1 | 1 | 1 |
| Treatment Week 4 | 28 ± 3 day | V4 | 1 | | | 1 | 1 | 1 | ✓ | | | | 1 | 1 | | | ✓ | ✓ | ✓ | ✓ |
| 6 | 42 ± 7 day | V5 | 1 | | | 1 | ✓ | | | | ✓• | | 1 | 1 | | | ✓ | 1 | 1 | ✓ |
| 8 (End treatment) | 56 ± 7 day | V6 | ✓ | | | 1 | 1 | | | | | | 1 | 1 | | | ✓ | ✓ | ✓ | ✓ |
| 10 | 70 ± 3 day | | | 1 | | 1 | 1 | | | | | | | 1 | | | | ✓ | ✓ | ✓ |
| 12 (SVR 4) | 84 ± 14 day | V7 | 1 | | | > | 1 | | | | ✓• | | | 1 | | | ✓ | 1 | 1 | 1 |
| 13 | 87 + 7 day | | | 1 | | | ✓ | | | | | | 1 | 1 | | | | | | |
| 16 (SVR 8) | 112 + 14 day | V8 | 1 | | | 1 | 1 | | ✓ | | | | 1 | 1 | | | ✓ | 1 | 1 | 1 |
| 20 (SVR-12) | 140 ±7 day | V9 | 1 | | | 1 | | 1 | ✓ | | | | 1 | 1 | | | | ✓ | ✓ | ✓ |
| 24 | 171 +14 day | | | 1 | | | | | | | | | 1 | 1 | | _ | | 1 | 1 | 1 |
| 28 | 196 ±7 day | | | 1 | | | | | | | | | | 1 | | | | 1 | 1 | 1 |
| 32 (SVR 24) | 224 ±7 day | | | 1 | | | | | | | | | | 1 | | | | 1 | 1 | 1 |
| 36 | 252 ±7 day | | | 1 | | | | | | | | | 1 | 1 | | | | 1 | 1 | 1 |
| 40 | 280 ±14 day | | | 1 | | | | | | | | | | 1 | | | | 1 | 1 | 1 |
| 52 | 365 ±14 day | V10 | 1 | | | 1 | | 1 | 1 | | | | 1 | 1 | | | ✓ | 1 | 1 | 1 |

<sup>\*</sup> CMP=comprehensive metabolic panel which includes basic metabolic panel and liver function tests \*\*As needed \$\delta\text{Viral Kinetics testing can be done anytime there is a standard of care blood draw \$\delta\text{If patients require the 16 weeks of therapy, the last 4 weeks would be the same as weeks 9-12 of therapy. If patients require only 8 weeks of therapy, then the lab test schedule will be modified to calculate \$\text{SVR 4, 8 and 12 based on end of therapy}\$

\[
\begin{array}{c}
\text{ONIVITY MEDICAL TO BE TO B

### 8.2.2. Blood sampling volumes

| Maximum Post-Transplant Blood Draw Totals | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Week<br>Post-KT | СВС | СМР | Tacrolimus | LFTs | HCV<br>RNA | HBV Core<br>Antibody | Viral Kinetics<br>(optional) | NS5A<br>Resistance | Blood Draw Total |
| 1 | 4 | 4.5 | 4 | 0 | 6 | 4 | 6 | 6 | 34.5 |
| 1 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 24.5 |
| 2 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 24.5 |
| 2 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 24.5 |
| 3 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 24.5 |
| 4 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 18.5 |
| 5 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 6 | 4 | 4.5 | 4 | 0 | 6 | 4 | 6 | 0 | 28.5 |
| 7 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 8 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 24.5 |
| 9 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 6 |
| 10 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 11 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 6 |
| 12 | 4 | 4.5 | 4 | 0 | 6 | 4 | 6 | 0 | 28.5 |
| 13 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 6 |
| 14 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 15 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 6 |
| 16 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 24.5 |
| 18 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 20 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 24.5 |
| 22 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 24 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 28 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 32 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 36 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 24.5 |
| 40 | 4 | 4.5 | 4 | 0 | 0 | 0 | 6 | 0 | 18.5 |
| 52 | 4 | 4.5 | 4 | 0 | 6 | 0 | 6 | 0 | 24.5 |
| Total | 92 | 103.5 | 92 | 0 | 84 | 12 | 162 | 6 | 551.5 |

<sup>♦</sup> There may be additional blood draws due to optional Viral Kinetics lab testing increasing the total sample volume.

#### 8.3. Subject retention and drug adherence

We will enforce subject retention in several ways. We will record extensive contact information for each subject at their enrollment in the trial. This will include home, work, and cellular telephone numbers. The research staff will call before each study visit to remind the subject to attend. We will also obtain contact information of a family member or friend so that we can contact him/her if the subject does not answer his/her regular phone number.

An adequate record of receipt, distribution, and return of all study drugs must be kept. Subject adherence with the treatment and protocol includes willingness to comply with all aspects of the protocol, and to have blood collected for all safety evaluations.

The research staff and physician will explain the importance of adherence with the study protocol at each subject contact. If a subject fails to comply with a study visit, the staff will contact him or her by telephone.

We have considered how to minimize non-adherence with therapy. We will strongly emphasize the importance of complying with the study drug treatment. Nonetheless, we will perform pill counts at visits and record episodes when medication is withheld for any reason. If a subject has a serious adverse event (SAE) (whether related to study drugs or not), we will continue to follow-up with the subject for study assessments to assist with safety monitoring and to avoid the problems introduced by missing data. The inclusion of such follow-up data will allow for analysis by intention-to-treat. If a study subject withdraws consent, he/she will no longer be followed.

### 9 Chapter 6: Assessment Of Efficacy And Outcome Measures

#### 9.1. Assessments of Efficacy

The primary aims of the study are to determine sustained virologic response rates (SVR) of open-label Zepatier, Mavyret, Epclusa or another appropriate antiviral treatment administered to HCV-negative patients with end-stage renal disease who receive a kidney transplant from an HCV-infected donor, leading to post-transplant denovo HCV infection.

#### 9.1.1. Sustained Virologic Response (SVR)

SVR will be based on the standard definition of SVR-12, defined as an undetectable HCV RNA in a subject's serum 12 weeks after completing treatment for HCV (12 weeks after the subject takes the last dose of Zepatier, Mavyret, Epclusa or another appropriate antiviral treatment).

#### 9.2. Secondary Outcome Measures

- To determine safety of administering Zepatier, Mavyret, Epclusa or another appropriate antiviral treatment to kidney transplant recipients who were previously HCV-negative, but developed denovo HCV after receiving a kidney transplant from an HCV-infected donor
- To determine 1-year graft survival rates of HCV-negative kidney transplant patients who receive a kidney transplant from an HCV-infected donor, including those who spontaneously clear HCV and those who receive open-label Zepatier, Mavyret, Epclusa or another appropriate antiviral treatment upon development of de-novo HCV.
- To evaluate rates of spontaneous clearance of HCV among HCV-negative patients who receive a kidney transplant from an HCV-infected donor.

#### 9.2.1. Safety

Subject safety and adverse events will be based in CTCAE Version 4 criteria, listed in Section 13, and will include adverse events and serious adverse events, related both to receipt of a kidney transplant from an HCV-positive donor among HCV-negative subjects with end-stage renal disease, and adverse events related to administration of Zepatier, Mavyret, Epclusa or another appropriate antiviral treatment.

#### 9.2.2. Graft Survival

Graft survival will be based on standardize United Network for Organ Sharing (UNOS) criteria, with a graft failure defined as subject death, re-transplantation, or chronic dialysis within the first year post-transplantation.

### 9.2.3. Spontaneous Clearance or Non-Transmission of HCV

Spontaneous clearance or non-transmission of HCV will be based on an undetectable HCV RNA level at post-transplant weeks 1-4 in the absence of treatment among HCV-negative subjects who receive a kidney transplant from a confirmed HCV-infected donor. Any subject who experiences spontaneous clearance of HCV or non-transmission of HCV will still be tested for HCV RNA at weeks 8, 16, and 28, to ensure that their levels are still undetectable.

### 10 CHAPTER 7: STATISTICAL CONSIDERATIONS

#### 10.1. Study Design

This open-label trial involves one primary and several secondary objectives. Post-transplant HCV status will be monitored, and patients will be treated with 8 to 12 weeks of therapy with Zepatier, Mavyret, Epclusa or another appropriate antiviral treatment, after which time, treatment will be complete, barring instances of treatment failure, which would require an additional course of therapy.\*

#### 10.2. Disposition of Subjects and Baseline Comparisons

Summaries of all subjects screened, recruited, and enrolled will be provided, according to the CONSORT guidelines. The treatment groups will be evaluated at baseline with respect to demographics and baseline measurements related to efficacy and safety without formal statistical testing.

#### 10.3. Analyses of Outcome Measures

The primary analysis will evaluate SVR-12 rates of HCV-negative kidney transplant recipients who receive a kidney from an HCV-infected donor and subsequently develop de-novo HCV. All patients will be assessed for toxicity and included in the safety analysis. This analysis will include summaries of the incidence and grade of toxicities. Patients will be evaluated for serious adverse events. Safety interim analyses will be performed and reported at each DSMB meeting.

#### 10.4. Missing Data and Dropouts

We will attempt to minimize missing data; however we have planned for its occurrence. For subjects lost to follow-up, we will use all of the information available until the end of follow-up. Subjects who withdraw consent will no longer be followed in this protocol. Patients will receive care from the patients' clinicians.

For patients lost to follow-up, we will use all the information available up to the time of loss to follow-up. For the primary end point, we will perform an analysis of completers only. We will also perform additional sensitivity analyses using imputation to assess the impact of missing data for the primary and secondary end points.

#### 10.5. Protocol Violations

Serious protocol deviations such as discontinuation of experimental treatment unrelated to adverse events (AEs) will be carefully recorded and regularly reviewed by co-Principal Investigators. Remedial changes in procedure will be recommended where feasible to reduce the incidence of such deviations. The causes and circumstances of all violations will be documented where known for purposes of future secondary analyses and interpretation. Because all primary analyses will be intent-to-treat, it is essential that violations be kept to a minimum, especially where it is possible to influence their rate of occurrence. A missed study visit will not be considered a protocol violation unless the study drug was scheduled to be dispensed at the visit, the subject did not have necessary labs done, or the subject has not been stable.

#### 10.6. Safety Analysis

All patients will be assessed for toxicity and included in the safety analysis. This analysis will include summaries of the incidence and grade of toxicities. Safety interim analyses will be performed at days 14, 30, 60, 90, 118, and 184, and will be reported at each DSMB meeting. SAEs will be evaluated by the DSMB.

### 11 CHAPTER 8: QUALITY CONTROL AND DATA HANDLING

#### 11.1. Personnel Training

Prior to enrolling the first subject in the study protocol, the PIs will ensure that the Investigator staff has completed appropriate training and that all documentation including IRB approval is completed and available. The purpose of training is to ensure that study personnel are carrying out the protocol in a consistent way and adhering to good clinical practice guidelines. Staff will have current Human Subjects Training Certification on file. Before enrollment begins, study staff who will perform the outcome assessments will be trained in all procedures, including completion of the REDCap database.

The co-PIs and research staff will constitute the first line of monitoring of the safety of the human participants. Surveillance for AEs will consist of questioning subjects about potential AEs at every study contact, having subjects report any AE to the study team, and having subjects undergo vital sign checks and physical exams during each study visit. Laboratories will be performed at selected visits and checked.

All study personnel are required to read the consent form, the protocol, and the IB.

#### 11.2. Data Quality

The co-PIs and research staff will perform continuous monitoring of data quality and completion of CRFs. Summary statistics from the screening logs will be sent to Merck quarterly or as requested. Finally, Merck staff reviews the reporting, documentation and follow-up of SAEs to assure that these events were handled according to required study procedures. All data on AEs and SAEs will be made available to the DSMB, as per the timeline outlined in the DSMB Charter.

#### 11.3. Audit and Inspection

Inspections may be carried out by regulatory health authority representatives [i.e., FDA] as well as the IRB.

#### 11.4. Archiving

Essential documents shall be archived safely and securely in such a way that ensures that they are readily available upon authorities' request. Patient (hospital) files will be archived according to local regulations and in accordance with the maximum period of time permitted by the hospital, institution or private practice.

### 12 Chapter 9: Participant Safety and Confidentiality

#### 12.1. Informed Consent and eConsent (i.e., remote consent)

Informed Consent will be obtained for enrollment from participants. For each consent process, whether inperson or by video conference, study personnel will discuss the details of the study, the risks and benefits, and the subject's rights and responsibilities if they choose to participate in the trial and their right to refuse to participate. It will be made clear that their clinical care will not be affected by their decision.

Each subject will have ample time and opportunity to ask questions and will be informed about the right to withdraw from the study at any time without any disadvantage and without having to provide reasons for this decision.

Only after the subject consents voluntarily and agrees to sign, in-person or electronically (eSign), the ICF and has done so, may he/she enter the study. Additionally, the investigator and other information provider (if any) will sign and date or digitally affirm the form. The subject will receive a paper or digital copy of the signed and dated form, as appropriate. All eConsents will adhere to current Office of Clinical Research approved procedures and regulations.

The signed informed consent statement is to remain in the investigator site file.

If the patient is not capable of providing a signature, a verbal statement of consent can also be given in the presence of an impartial witness (independent of the investigator). This is to be documented by a signature from the informing physician as well as by a signature from the witness.

The ICF and any other written information provided to subjects / legal representatives or proxy consenters will be revised whenever important new information becomes available that may be relevant to the subject's consent, or there is an amendment to the protocol that necessitates a change to the content of the subject information and / or the ICF. The investigator will inform the subject / legal representative or proxy consenter of changes in a timely manner and will ask the subject to confirm his/her participation in the study by signing, inperson or electronically (eSign), the revised ICF. Any revised ICF and written information must receive the IEC/IRB's approval in advance of use.

#### 12.2. Institutional Review Board Process

Study staff will obtain IRB approval before any study procedures are initiated.

#### 12.3. Insurance

The kidney transplant itself will be paid for by subjects' insurance carriers, and does not require any additional pre-authorization because of the potential to receive a kidney from a hepatitis C-positive donor. The costs of all visits and tests described above will be billed to the insurance carrier, except for: 1) the blood draw for research purposes (which includes the hepatitis C genotype test, which is based on a laboratory-developed test using materials purchased from the commercial entity that developed this test, and will be paid for by the research team), 2) the study drug Zepatier in the event of infections with genotype 1 or genotype 4 HCV, which will be provided by Merck, and 3) other antiviral therapies for infections with HCV that are neither genotype 1 nor genotype 4; these therapies will be provided by HUP until such time that the subject's insurance provides coverage for the drug. In the event that the subject's insurance denies coverage for the treatment, HUP will provide the full course of appropriate HCV therapy as well as a second treatment course of antiviral therapy for HCV if the first treatment fails.

Subjects are still responsible for any deductibles or applicable co-pays for routine office visits, blood work and scans (except for the liver Fibroscans listed above). We do not expect subjects to have health insurance coverage/payment issues due to becoming infected with hepatitis C, per se, and the study is designed so subjects do not require additional study visits post-transplant, provided there are no adverse events.

#### 12.4. Laboratory Values

The following clinical laboratory tests will be measured and repeated at time points specified in schedule of procedures (section 8.2.1) and as clinically indicated.

#### 12.4.1. Chemistry

- Hepatic function panel including alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total and direct bilirubin, and albumin.
- Basic metabolic panel including BUN and creatinine.

#### 12.4.2. Serum virologic testing

- HCV RNA (with Genotyping per protocol)
- Hepatitis B surface antigen
- HIV antibody testing.
- HBV Core Antibody (as needed)

#### 12.4.3. Pregnancy Testing

Blood and urine pregnancy tests will be performed (as appropriate) per the schedule of procedures (section 5.2).

#### 12.4.4. Hepatitis C Viral Kinetics

Each time standard of care laboratories are drawn, subjects may have one additional purple -top tube drawn (4cc of blood). This blood test is considered optional. The research coordinator will process the tube and store it in a -80° freezer in the Perelman Center for Advanced Medicine 7<sup>th</sup> Floor Gastroenterology Research Office. Each month, these tubes will be shipped to Abbott Pharmaceuticals so they can test for HCV antibodies, HCV core antigen, and HCV RNA. These additional tests will be included in the informed consent process for all subjects. Abbott will perform these tests free of charge to University of Pennsylvania once both are able to reach a Material Transfer Agreement (MTA).

#### 12.5. Zepatier Related Laboratory Abnormalities and Drug Interactions

**Laboratory Abnormalities** 

The following laboratory abnormalities were observed in studies done with Zepatier:

Late elevations in aminotransferase levels greater than 5 times the upper limit of normal generally occurred in around 1-3% of patients in previous Zepatier clinical trials; these increases were rarely associated with hyperbilirubinemia. These abnormalities were reversible and had no major clinical consequences.

Effects of Zepatier on antiretrovirals:

Atazanavir/ritonavir 300/100mg co-administered with MK-5172 200mg daily somewhat increased atazanavir exposure (AUC increased 43%, Cmax increased 12%, C24 increased 23%). Co-administration of these medications is not recommended.
- Darunivir/ritonavir 600/100 mg co-administered with MK-5172 200 mg was not significantly altered by either MK-5172 or MK-8742. However, due to DRV/r effects on Zepatier exposure, co-administration is not recommended.
- Efavirenz was not significantly impacted when co-administered with Zepatier, though it may negatively impact Zepatier exposure.
- Lopinavir/ritonavir exposures were not significantly impacted when co-administered with Zepatier. However, due to LPV/r effects on Zepatier exposure, co-administration is not recommended.

### Effect of Antiretrovirals on Zepatier:

- Atazanavir/ritonavir 300/100mg co-administered with MK-5172 200mg significantly increased exposure
  of MK-5172 (AUC increased 10.58-fold, Cmax increased 6.24-fold, and C24 increased 11.6-fold). These
  findings were similar when ATV/r was combined with 50mg MK-8742. MK-8742 AUC geometric mean
  ratio (GMR) was 4.76, probably due to ATV/r CYP3A4/Pgp inhibition and possible inhibition of OATPmediated disposition of MK-8742. Co-administration of these medications is not recommended.
- Exposures of MK-5172 were significantly increased when MK-5172 200 mg was co-administered with darunavir/ritonavir 600/100 mg daily. MK-5172 AUC increased 7.5-fold, Cmax increased 5.27-fold, and C24 increased 8-fold. MK-8742 exposures were also significantly increased when combined with DRV/r 600/100 mg daily. MK-8742 AUC GMR following co-administration was 1.66. This increase is likely caused by CYP3A4/Pgp inhibition by DRV/r and possibly inhibition of OATP-mediated disposition of MK-8742. For these reasons, co-administration of Zepatier and DVR/r is not recommended.
- Efavirenz 600mg co-administration with MK-5172 200 mg decreased MK-5172 AUC by 84%, most likely due to CYP3A4 induction. The same dose EFV combined with MK-5172 50 mg also decreased MK-8742 AUC 54% for the same reasons. Co-administration of these medications may cause sub-therapeutic MK-5172 exposure.
- Lopinavir/ritonavir 400/100 mg co-administered with MK-5172 200 mg significantly increased MK-5172 exposure. MK-5172 AUC increased 12.86-fold, Cmax increase 7.31-fold, and C24 increased 21.7-fold. When the same dose of LPV/r was administered with MK-8742 50 mg, MK-8742 AUC GMR was increased to 3.71. LPV/r likely impacts MK-8742 exposures due to CYP3A4/Pgp inhibition and possible inhibition of OATP-mediated disposition. Co-administration of these medications is not recommended.

#### Effect of Zepatier on Other Drugs:

- Rosuvastatin 10 mg co-administered with Zepatier 200/50 mg increased rosuvastatin exposure.
   Rosuvastatin AUC and Cmax were increased 59% and 325% respectively when exposed to MK-5172 alone and 126% and 449% when exposed to the combined Zepatier pill. The most likely cause of the increase is pre-systemic inhibition of rosuvastatin efflux in the liver and/or gut due to BCRP inhibition. Clinicians may want to avoid co-administration of Zepatier and rosuvastatin.
- Midazolam 2 mg/mL combined with multi-dose MK-5172 200 mg daily decreased midazolam AUC to 34%. MK-5172 is likely a weak CYP3A4 inhibitor.
- Multiple oral doses of rifampin did not significantly affect MK-5172 AUC, but reduced C24h by 85%. This
  decrease was presumably due to the combined effect of OATP inhibition and CYP3A4/Pgp induction by
  chronic rifampin administration. Clinicians should avoid co-administration of these medications until
  further data becomes available.

#### Effect of Other Drugs on Zepatier:

 Rosuvastatin 10 mg co-administered with Zepatier 200/50 mg did not significantly alter MK-5172/8742 exposure. However, due to Zepatier effects on rosuvastatin exposure, clinicians may wish to avoid co-administration.

- Ketoconazole (CYP3A4 and P-gp inhibitor) approximately tripled MK-5172 AUC. In healthy male subjects taking 400 mg multi-dose ketoconazole, MK-8742 AUC increased by 31%.
- Combining MK-5172 200 mg and a single dose of 600 mg IV rifampin caused a 12.6-fold increase in MK-5172 AUC, compared to an 8.35-fold increase with a single dose of oral rifampin 600 mg. This is likely due to P-gp and OATP inhibition by rifampin. Clinicians should avoid co-administration of these medications until further data becomes available.

### 12.6. Mavyret Related Laboratory Abnormalities and Drug Interactions

Subjects must be able to safely discontinue any prohibited medications or supplements listed in the Table prior to the first dose of Mavyret and not use these during the entire Treatment Period and for 2 weeks following discontinuation of study drugs.

## **Table: Prohibited Medications and Supplements**

### **Medication or Supplement Name**

- Red yeast rice (monacolin K), St. John's Wort
- Ethinyl estradiol
- Atorvastatin, lovastatin, simvastatin
- Carbamazepine, phenytoin, pentobarbital, phenobarbital, primidone, rifabutin, rifampin
- Astemizole, cisapride, terfenadine

Use of high dose (0.035mg) ethinyl estradiol containing oral contraceptives with Mavyret combination was associated with asymptomatic ALT increases (one Grade 3, and one Grade 2) without concurrent bilirubin increases in 2 healthy female subjects. Therefore hormonal contraceptives (including oral, topical [including vaginal rings], injectable or implantable varieties) containing any ethinyl estradiol may not be used from 2 weeks prior to the first dose of study drug until 2 weeks after the end of study drug dosing. Progestin-only contraceptives, such as those containing norethindrone, desogestrel, or levonorgestrel, without ethinyl estradiol, may be used with Mavyret. Post-menopausal hormone replacement therapy, such as with esterified or conjugated estrogens, i.e., not containing ethinyl estradiol, may be used with Mavyret at the discretion of the Investigator.

Mavyret may be initiated in subjects receiving cyclosporine ≤100 mg per day. Concomitant administration of Mavyret with cyclosporine doses of greater than 100mg per day is <u>not</u> recommended.

### 12.7. Epclusa Related Laboratory Abnormalities and Drug Interactions

Effects of Epclusa on Other Drugs:

• Velpatasvir is an inhibitor of drug transporters P-gp, breast cancer resistance protein (BCRP), OATP1B1, OATP1B3, and OATP2B1. Coadministration of Epclusa with drugs that are substrates of these transporters may increase the exposure of such drugs.

• Fluctuations in INR values may occur in patients receiving warfarin concomitant with HCV treatment, including treatment with Epclusa. Frequent monitoring of INR values is recommended during treatment and post-treatment follow-up.

## Effects of Other Drugs on Epclusa:

- Sofosbuvir and velpatasvir are substrates of drug transporters P-gp and BCRP while GS-331007 (the
  predominant circulating metabolite of sofosbuvir) is not. In vitro, slow metabolic turnover of velpatasvir
  by CYP2B6, CYP2C8, and CYP3A4 was observed.
- Drugs that are inducers of P-gp and/or moderate to potent inducers of CYP2B6, CYP2C8, or CYP3A4 (e.g., rifampin, St. John's wort, carbamazepine) may decrease plasma concentrations of sofosbuvir and/or velpatasvir, leading to reduced therapeutic effect of Epclusa. The use of these agents with Epclusa is not recommended. Epclusa may be coadministered with P-gp, BCRP, and CYP inhibitors.

Established and Potentially Significant Drug Interactions:

• See Table on next page.

| Concomitant Drug Class: Drug<br>Name | Effect on<br>Concentration <sup>b</sup> | Clinical Effect/Recommendation |
|---|---|---|
| Acid Reducing Agents: | ↓ velpatasvir | Velpatasvir solubility decreases as pH increases. Drugs that increase gastric pH are expected to decrease concentration of velpatasvir. |
| Antacids (e.g., aluminum and magnesium hydroxide) | | Separate antacid and EPCLUSA administration by 4 hours. |
| H <sub>2</sub> -receptor antagonists <sup>c</sup> (e.g., famotidine) | | H <sub>2</sub> -receptor antagonists may be administered simultaneously with or 12 hours apart from EPCLUSA at a dose that does not exceed doses comparable to famotidine 40 mg twice daily. |
| Proton-pump inhibitors <sup>C</sup><br>(e.g., omeprazole) | | Coadministration of omeprazole or other proton-pump inhibitors is not recommended. If it is considered medically necessary to coadminister, EPCLUSA should be administered with food and taken 4 hours before omeprazole 20 mg. Use with other proton pump- inhibitors has not been studied. |
| Antiarrhythmics:<br>amiodarone | Effect on<br>amiodarone,<br>sofosbuvir, and<br>velpatasvir<br>concentrations<br>unknown | Coadministration of amiodarone with EPCLUSA may result in serious symptomatic bradycardia. The mechanism of this effect is unknown. Coadministration of amiodarone with EPCLUSA is not recommended; if coadministration is required, cardiac monitoring is recommended [see Warnings and Precautions (5.1) and Adverse Reactions (6.2)]. |
| digoxin <sup>©</sup> | ↑ digoxin | Therapeutic concentration monitoring of digoxin is recommended when coadministered with EPCLUSA. Refer to digoxin prescribing information for monitoring and dose modification recommendations for concentration increases of less than 50%. |
| Anticancers: topotecan | ↑ topotecan | Coadministration is not recommended. |
| Anticonvulsants: carbamazepine phenytoin phenobarbital oxcarbazepine | ↓ sofosbuvir<br>↓ velpatasvir | Coadministration is not recommended. |
| Antimycobacterials:<br>rifabutin rifampin <sup>C</sup><br>rifapentine | ↓ sofosbuvir<br>↓ velpatasvir | Coadministration is not recommended. |
| HIV Antiretrovirals: | | To |
| eravirenz | ↓ velpatasvir | Coadministration of EPCLUSA with efavirenz-containing regimens is not recommended. |
| Regimens containing tenofovir<br>DF | ↑ tenofovir | Monitor for tenofovir-associated adverse reactions in patients receiving EPCLUSA concomitantly with a regimen containing tenofovir DF. Refer to the prescribing information of the tenofovir DF-containing product for recommendations on renal monitoring. |
| tipranavir/ritonavir | ↓ sofosbuvir<br>↓ velpatasvir | Coadministration is not recommended. |
| Herbal Supplements: | ↓ sofosbuvir | Coadministration is not recommended. |
| St. John's wort (Hypericum perforatum) | ↓ velpatasvir | |
| HMG-CoA Reductase Inhibitors: rosuvastatin <sup>C</sup> | ↑ rosuvastatin | Coadministration of EPCLUSA with rosuvastatin may significantly increase the concentration of rosuvastatin, which is associated with increased risk of myopathy, including rhabdomyolysis. Rosuvastatin may be administered with EPCLUSA at a dose that does not exceed 10 mg. |
| atorvastatin | ↑ atorvastatin | Coadministration of EPCLUSA with atorvastatin is expected to increase the concentrations of atorvastatin, which is associated with increased risk of myopathy, including rhabdomyolysis. Monitor closely for HMG- CoA reductase inhibitor-associated adverse reactions, such as myopathy and rhabdomyolysis. |

DF = disoproxil fumarate

a. This table is not all inc

b. ↓ = decrease, ↑ = increase

c. These interactions have been studied in healthy adults.

#### 12.8. Other Events

We will not discontinue study drug for clinical events not thought to be serious drug-related AEs. For example, a hospitalization for clinical worsening may or may not result in cessation of trial participation. Such events could result in missing data for primary and secondary endpoints, comprising the integrity of the analysis. This trial does prohibit certain therapies, thus there may be a reason to stop study drug participation under such circumstances. Even if subjects are withdrawn from the study drug, outcome assessments will continue, allowing analysis by intent-to-treat.

### 12.9. Safety and Adverse Events

#### 12.9.1. Definitions

**Adverse event (AE)**: Any untoward medical occurrence associated with the protocol procedures, whether or not considered product or process related. Any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. Inter-current illnesses or injuries should be regarded as AEs. Abnormal results of diagnostic procedures are considered to be AEs if the abnormality:

- results in study withdrawal
- is associated with a serious AE
- is associated with clinical signs or symptoms
- leads to additional treatment or to further diagnostic tests
- is considered by the investigator to be of clinical significance

**Serious adverse event (SAE):** Adverse events are classified as serious or non-serious. A **serious adverse event** is any AE that is:

- fatal
- life-threatening
- requires or prolongs hospital stay
- results in persistent or significant disability or incapacity
- a congenital anomaly or birth defect
- an important medical event

Important medical events are those that may not be immediately life threatening, but are clearly of major clinical significance. They may jeopardize the subject, and may require intervention to prevent one of the other serious outcomes noted above. For example, drug overdose or abuse, a seizure that did not result in in-subject hospitalization or intensive treatment of bronchospasm in an emergency department would typically be considered serious.

All AEs that do not meet any of the criteria for serious should be regarded as non-serious AEs.

**Suspected adverse reaction:** Any adverse event for which there is a reasonable possibility that the drug/investigational product caused the adverse event. For reporting purposes, "reasonable possibility" means there is evidence to suggest a causal relationship between the drug/investigational product and the adverse event.

**Unanticipated Adverse Device Effect (ADE):** is any serious adverse effect on health or safety, or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application, or any

other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

### 12.9.2. Classifying Adverse Events

#### Severity

The intensity of the AE is classified according to the CTCAEv4.0.<sup>23</sup> Grade refers to the severity (intensity) of the AE:

- **CTCAEv4 Grade 1**: **mild**; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention is not indicated.
- **CTCAEv4 Grade 2**: **moderate**; minimal, local, or noninvasive intervention is indicated; limiting to ageappropriate instrumental activities of daily living (ADL; instrumental ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.).
- **CTCAEv4 Grade 3**: **severe** or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization is indicated; disabling; limiting to self-care ADL (self-care ADL refers to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden).

CTCAEv4 Grade 4: life-threatening consequences; urgent intervention is indicated.

CTCAEv4 Grade 5: death due to an AE.

#### **Expectedness**

AEs must be assessed as to whether they were expected to occur or were unexpected, meaning not anticipated based on current knowledge found in the protocol, investigator brochure, product insert, or label.

**Expected:** an AE/ADE known to be associated with the intervention or condition under study.

**Unexpected:** an AE/ADE for which the nature or severity is not consistent with information about the condition under study or intervention in the protocol, consent form, product brochure, or investigator brochure.

OHRP defines an **unexpected AE** as any AE occurring in one or more subjects participating in a research protocol, the nature, severity, or frequency of which is **not** consistent with either:

- 1) the known or foreseeable risk of AEs associated with the procedures involved in the research that are described in a) the protocol-related documents, such as the IRB-approved research protocol, any applicable investigator brochure, and the current IRB-approved informed consent document, and b) other relevant sources of information, such as product labeling and package inserts; or
- 2) the expected natural progression of any underlying disease, disorder, or condition of the subject(s) experiencing the AE and the subject's predisposing risk factor profile for the AE.

#### Relatedness

- 1) Definite: the AE/ADE is clearly related to the research procedures
- 2) **Probably:** the AE/ADE is likely related to the research procedures
- **3) Possible:** the AE/ADE may be related to the research procedures
- **4) Unlikely:** the AE/ADE is doubtfully related to the research procedures
- **5) Unrelated:** the AE/ADE is clearly not related to the research procedures

For each identified AE/ADE, an entry on the AE/ADE form will be completed. Reporting procedures should be started immediately upon learning of a SAE/ADE.

#### 12.9.3. Interpretation of Definitions

### **AE Reporting Period**

The study period during which AEs must be reported is normally defined as the time of consent to the end of the study treatment follow-up. However, for this study, the AE reporting period will be divided based on the three phases of the study.

a. Screening phase: When all screening tests have been done, we will assess for any AEs related to the screening tests at the time of communication with the subject about whether he/she is official eligible or ineligible for the study.

**Preexisting Condition:** A preexisting condition is one that is present at the start of the study. A preexisting condition should be recorded as an AE if the frequency, intensity, or the character of the condition worsens during the study period.

- **b. Waitlist phase**: We will only capture AEs that are pertinent to the study. Specifically the following will be captured:
  - 1. Patient death,
  - 2. Patient develops a condition that would exclude them from the study,
  - 3. Patient is de-listed (taken off the kidney transplant waitlist),
  - 4. Patient is made inactive on the transplant waitlist,
  - **5.** Patient is transplanted with a non-HCV kidney.

In order to ascertain these events, we will review the patient's medical record once a month, and will contact the patient (by phone, e-mail, or in-person) every 6-8 weeks.

- **c. Post-transplant phase**: All AEs will be assessed at every clinic visit when the subject is seen by a member of the study team.
- **d. Post-study:** At the last scheduled visit, the investigator will instruct each subject to report any subsequent event(s) that the subject, or the subject's personal physician, believes might reasonably be related to participation in this study.

All unresolved AEs considered possibly, probably or definitely related to the study drug should be followed by the investigator until the events are resolved, the subject is lost to follow-up, or the AE is otherwise explained. The investigator will notify the IRB of any death or AE occurring at any time after a subject has discontinued or terminated study participation that may reasonably be related to this study. The IRB will also be notified if the investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject that has participated in this study.

### General Physical Examination Findings (screening, post-transplant, and post-study phases)

At screening, any clinically significant abnormality should be recorded as a preexisting condition. At the end of the study, any new clinically significant findings/abnormalities that meet the definition of an AE must also be recorded and documented as an AE.

### Abnormal Laboratory Values (post-transplant, and post-study phases)

A clinical laboratory abnormality should be documented as an AE if any one of the following conditions is met:

- The laboratory abnormality is considered clinically significant by the local PI and is not otherwise refuted by a repeat test to confirm the abnormality
- The abnormality suggests a disease and/or organ toxicity
- The abnormality is of a degree that requires active management; e.g. change of dose, discontinuation of the drug, more frequent follow-up assessments, further diagnostic investigation, etc.

### Hospitalization, Prolonged Hospitalization or Surgery (post-transplant and post-study phase)

Any AE that results in hospitalization or prolonged hospitalization should be documented and reported as a serious AE unless specifically instructed otherwise in this protocol, with the exception of hospitalization at the time of a kidney offer and/or kidney transplant. Any condition responsible for surgery should be documented as an AE if the condition meets the criteria for and AE.

Neither the condition, hospitalization, prolonged hospitalization, nor surgery are reported as an AE in the following circumstances:

- Hospitalization or prolonged hospitalization for diagnostic or elective surgical procedures for a
  preexisting condition. Surgery should *not* be reported as an outcome of an AE if the purpose of the
  surgery was elective or diagnostic and the outcome was uneventful.
- Hospitalization or prolonged hospitalization for therapy of the target disease of the study, unless it is a worsening or increase in frequency of hospital admissions as judged by the clinical investigator.

### 12.9.4. Reporting Procedures for Unanticipated Problems, Adverse Events, and Adverse Device Effects

Principal investigators should notify the local IRB, in an expedited manner, of those events related to study participation that are unforeseen and indicate that participants or others are at increased risk of harm. Researchers should submit reports of the following problems:

Any AE/ADE or UP (regardless of whether the event is serious or non-serious, on-site or off-site) that occurs any time during or after the research study, which in the opinion of the principal investigator is:

Unexpected (An event is "unexpected" when its specificity and severity are not accurately reflected in the protocol-related documents, such as the IRB-approved research protocol, any applicable investigator brochure, and the current IRB-approved informed consent document and other relevant sources of information, such as product labeling and package inserts.)

#### **AND**

Related to the research procedures (An event is "related to the research procedures" if in the opinion of the principal investigator, the event was more likely than not to be caused by the research procedures.)

#### **AND**

Suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

Additionally, all adverse events/adverse device effects shall be documented by the PI team and assessed. All Serious Adverse Events will be forwarded to **Merck Worldwide Product Safety.** 

| What Event is Reported | By Whom is Event<br>Reported | To Whom is Event<br>Reported | When is Event Reported |
|---|---|---|---|
| Fatal unexpected, suspected serious adverse event | Investigator | Local IRB | Within <b>24 hours</b> of initial receipt of information |

| (SAE/ADE – death that is unexpected and poss/prob/def related to the research) | | | |
|---|---|---|---|
| Life-threatening unexpected, suspected serious adverse reactions (SAE/ADE- life-threatening, | Investigator | Local IRB | |
| unexpected, poss/prob/def related to the research) | | | Within <b>3 calendar days</b> of |
| Non-fatal, non-life-threatening unexpected, suspected serious adverse reactions | | | initial receipt of information |
| (SAE/ADE – unexpected, poss/prob/def related, non-life-threatening hospitalization, prolonged hospitalization, disability/incapacity/birth defects, important medical event) | Investigator | Local IRB | |
| Unanticipated Problem that is not an SAE (AE/ADE or non-AE, unexpected, poss/prob/def related and suggests greater risk of harm) e.g. Development of moderate hypersomnia that resolve after discontinuing drug. This AE/ADE although not-serious, is not listed as an expected event in the consent. Thus it is an AE that is unexpected, possibly related (resolved after a prince) | Investigator | Local IRB | Within <b>10 calendar days</b> of initial receipt of information |
| possibly related (resolved after coming off drug), and places subject(s) at greater risk of harm than previously known | | | |

## 12.9.4.1. Reporting Process

UPs posing risks to subjects or others as noted above will be reported to the local IRB using a Medwatch or CIOMS report of the event (including a description of the event with information regarding its fulfillment of the above criteria, follow-up/resolution and need for revision to consent form and/or other study documentation) will be completed

All Serious Adverse Events, regardless of causal relationship to the investigational product, will be forwarded to **Merck Worldwide Product Safety** via fax (**215-993-1220**) within 2 working days of the investigator becoming aware of the event and no later than 3 calendar days.

The Principal Investigator is expected to provide as much of the following information:

- · Protocol name and number
- Subject identifiers
- · Demographic data
- Nature of the event
- Severity of the event
- · Probable relationship (causality) of AE to study procedure
- Date and time of AE onset
- · Date and time of AE resolution, if available
- · Concomitant medications that the participant was taking for an underlying medical condition or disease and the therapeutic agents used for the treatment of the adverse event
  - Clinical assessment of participant conducted at time of SAE/AE
  - Results of any laboratory and/or diagnostic procedures, and treatment
  - Follow-up plan
  - Outcome
  - Autopsy findings (if appropriate)

The Principal Investigator will provide details about the AE/ADE as they become available. If additional information cannot be obtained for whatever reason, this will be documented. The Principal Investigator should inform the IRB when no other information is expected. The Principal Investigator should provide the IRB with a logical, complete, and accurate narrative description of the SAE based upon the above information.

The Principal Investigator should promptly determine an assessment of causality.

The IRB determines if any corrective actions should be initiated as a result of any known specific or collective SAE/AE(s) and inform the principal investigator of the corrective action (e.g., revision of informed consent form, protocol, CRF).

The Principal Investigator/designee should keep originals or photocopies of all relevant documentation, including facsimile confirmations, and file them in the participant's file.

The Principal Investigator should ensure that all routine AE(s) are reported as part of the periodic or annual reporting requirements to the IRB of record.

The Principal Investigator should file copies of all correspondence with the IRB in the appropriate section of the Regulatory Master File or site study file.

### **Other Reportable Events:**

The following events are also reportable to the IRB:

- Any adverse experience that, even without detailed analysis, represents an unexpected SAE that is rare in the absence of drug exposure (such as agranulocytosis, hepatic necrosis).
- Any AE that would cause a modification to the investigators brochure, protocol or ICF, or would prompt other action by the IRB to assure protection of human subjects.

- Information that indicates a change to the risks or potential benefits of the research, in terms of severity or frequency. For example:
  - An interim analysis indicates that participants have a lower rate of response to treatment than initially expected.
  - Safety monitoring indicates that a particular side effect is more severe, or more frequent than initially expected.
  - A paper is published from another study that shows that an arm of your research study is of no therapeutic value.
- Breach of confidentiality
- Change to the protocol taken without prior IRB review to eliminate apparent immediate hazard to a research participant.
- Incarceration of a participant when the research was not previously approved under Subpart C and the investigator believes it is in the best interest of the subject to remain on the study.
- Complaint of a participant when the complaint indicates unexpected risks or the complaint cannot be resolved by the research team.
- Protocol violation (meaning an accidental or unintentional deviation from the IRB approved protocol) that in the opinion of the investigator placed one or more participants at increased risk, or affects the rights or welfare of subjects.

**Unanticipated Problem Involving Risks to Subjects or Others (UPRSO):** Any incident, experience, or outcome that meets **all** of the following criteria:

- 1) Unexpected (in terms of nature, severity, or frequency) given a) the research procedures that are described in the protocol-related documents, such as the IRB-approved research protocol, informed consent document, or investigators brochure; and b) the characteristics of the subject population being studied;
- 2) Related or possibly related to participation in the research (possibly related to participation in the research means there is a reasonable possibility that the AE, experience, or outcome may have been caused by the procedures involved in the research.); and
- 3) Suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

### 12.10. Subject Withdrawal

A subject has the right to withdraw from the study entirely at any time for any reason without prejudice to future medical care by the investigator or other physician. The investigator also has the right to withdraw subjects from the study in the event of concurrent illness, AEs, or other reasons deemed to be in the subject's best interest.

Subjects must be withdrawn from the trial (treatment and procedures) for the following reasons:

- Subject withdraws consent for study treatment and study procedures. A subject must be removed from
  the trial at his/her own request or at the request of his/her legally acceptable representative. At any
  time during the trial and without giving reasons, a subject may decline to participate further. The
  subject will not suffer any disadvantage as a result.
- Subject becomes pregnant while undergoing treatment—therapy will be stopped as there are no human safety data of the study drugs during pregnancy. There are no adequate and well-controlled

studies with the study drugs in pregnant women. No effects on embryo-fetal development were observed in rats or rabbits at grazoprevir or elbasvir exposures higher than exposures in humans at the recommended clinical dose. Because animal reproduction studies are not always predictive of human response, DAAs should be used during pregnancy only if the potential benefit justifies the potential risk to the fetus. Because the transmission rates of HCV from mother to fetus are very small, and HCV can be treated after pregnancy and delivery, therapy will not be continued during pregnancy. Patients will continue with the regularly scheduled study visits, but will not be eligible to receive continued therapy.

- Subject develops a condition that it is life threatening or any other significant risk as judged by the Investigators. Patients will not receive study drug, but will continue with study visits as scheduled.
- Zepatier, Mavyret, Epclusa, or other appropriate antiviral treatment is no longer produced by the company, or if a decision is made to stop the study patients will not receive study drug, but will continue with study visits as scheduled.

Any subject removed from the trial will remain under medical supervision until discharge or transfer is medically acceptable.

In all cases, the reason for withdrawal must be recorded in the CRF and in the subject's medical records.

In order to preserve the integrity of the intention-to-treat analysis, even if the subject is withdrawn from the treatment portion of the protocol (either due to subject, physician, or investigator decision), it is imperative to continue with the scheduled follow-up assessments both for the safety of the subject and for completeness of data collection. This will be explained to potential subjects at the time of informed consent. The importance of adherence with study visits will be reinforced throughout the trial. If the treatment is permanently withdrawn, the subject will return to the center for safety assessment (history, physical examination, and clinical laboratories, if necessary).

#### 12.11. Confidentiality of Study Data

Information about study subjects will be kept confidential and managed according to the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Those regulations require a signed subject authorization informing the subject of the following:

- What protected health information (PHI) will be collected from subjects in this study
- Who will have access to that information and why
- Who will use or disclose that information
- The rights of a research subject to revoke their authorization for use of their PHI

In the event that a subject revokes authorization to collect or use PHI, the investigator, by regulation, retains the ability to use all information collected prior to the revocation of subject authorization. For subjects that have revoked authorization to collect or use PHI, attempts should be made to obtain permission to collect at least vital status (i.e., that the subject is alive) at the end of their scheduled study period.

Should direct access to medical records require a waiver or authorization separate from the subject's statement of informed consent, it is the responsibility of the Investigator to obtain such permission in writing from the appropriate individual.

#### 12.12. Potential Risks

### 12.12.1. Risks of Study Procedures

There are several areas of potential risk in this study. We will obtain several blood samples from each subject. There is a risk of bruising, hematoma, and infection after phlebotomy, which are possible but not considered serious AEs. Fainting may occur, which is unlikely but considered a serious AE. The removal of <70 cc of blood every 1-4 weeks during the 40-week post-transplant period is a potential risk; however this amount is routinely taken from subjects for clinical indications without adverse effect. Study medications will be delayed until after phlebotomy on each study day.

Because we may store subjects' blood samples, there may be confidentiality risks associated with the storage and analysis of those samples or the information resulting from the analysis of those samples. Samples may be used for genetic testing. Under some circumstances, it can be a risk for genetic information to be known. To help ensure confidentiality, samples will be coded and stored in a secured facility. While situations cannot be foreseen where potentially sensitive genetic information is revealed or where people who should not have this information could obtain it (representing a loss of confidentiality), however, it is possible that presently unforeseen situations may arise where this could happen.

The risk of undergoing screening includes potential identification of new health problems that subjects were unaware of. If we discover new health problems, we will answer subjects' questions and try to arrange appropriate treatment if any is needed. If new health problems are discovered, it is possible that subjects would not be able to enter this study. It is also possible that subjects would no longer be eligible for kidney transplantation based on the results.

The risks associated with an echocardiogram are often none or include mild skin irritation or rash at the site of electrode placement.

The risks associated with a Fibroscan are that the probe used on the abdomen during the Fibroscan may lead to mild soreness in the area for about a day.

The risks of kidney transplant surgery include blood loss, infections, and deep vein thrombosis. There are also risks related to immunosuppression and standard anti-infective therapy.

The risks of any transplant include primary graft non-function, delayed graft function, acute rejection, and death. Re-admissions within 30 days after a kidney transplant are expected in approximately 40% of patients.

There may also be a small risk of developing Focal and Segmental Glomerulosclerosis (FSGS) after receiving a kidney from HCV positive donor. However, this condition can also develop in patients who do not have HCV. After transplant, we will monitor all patients for FSGS and similar conditions.

#### 12.12.2. Risk of Genotyping Failure

There is a risk of failure of the Genotyping LDT in that no result is obtained. In that case, the investigators will use their judgment to select the most appropriate empirical treatment regimen.

There is also a risk of the Genotyping LDT giving an incorrect genotype. The risk to the recipient participant, in this event, is that they receive the transplant, but are possibly unable to be adequately treated for HCV positivity. Failure of the LDT to give an accurate genotype could be due to a mixed infection (e.g. genotype 1 and 2) or HCV genotype 4f infection in the donor sample.

#### 12.12.3. Risk of NS5a Drug Resistance Test Failure

The potential risks of the NS5a resistance testing are false negative and false positive test results. The risk of a false negative test result would be if the test does not report any one of the four pertinent polymorphisms, even though they are present (the presence of which would be rare). In this case, the patient would receive only 12 weeks of Zepatier (rather than 16 weeks of Zepatier + renal-dosed Ribavirin), and potentially fail first-line therapy, requiring second-line therapy.

A false positive result is less likely to happen than a false negative result. The risk of a false positive test result would be if the test reports a polymorphism when the subject does not have one. Hence, the subject would be exposed to Zepatier for 4 weeks longer than needed as well as Ribavirin, and potentially experiencing the products' side effects.

### 12.12.4. Risk of Study Drugs

#### Zepatier

In subjects receiving Zepatier for 12 weeks, the most commonly reported adverse reactions of all intensity (greater than or equal to 5% in placebo-controlled trials) were fatigue, headache, and nausea. In subjects receiving Zepatier with ribavirin for 16 weeks, the most commonly reported adverse reactions of moderate or severe intensity (greater than or equal to 5%) were anemia and headache. <sup>24-26</sup>The greatest risk is failure to achieve SVR12 after treatment with Zepatier, leading to chronic HCV.

There is a risk of fetal harm and birth defects should any woman taking Zepatier become pregnant while on the drug. <sup>24-26</sup> Due to the age of the participants, this is a small risk, as all will be over 30 and few are likely to become pregnant. However, to mitigate this risk, all pre-menopausal women with a uterus will be screened for pregnancy before enrollment and instructed to use a highly effective form of birth control (e.g. abstinence, intrauterine device, etc.). Highly effective forms of birth control will be defined by the Mycophenolate Risk Evaluation and Mitigation Strategy (REMS), a standard protocol used for post-transplant patients at Penn being treated with Mycophenolate.

#### Sovaldi (Sofosbuvir)

The most common adverse events (incidence greater than or equal to 20%, all grades) observed with Sovaldi in combination with ribavirin were fatigue and headache. The most common adverse events observed with Sovaldi in combination with peginterferon alfa and ribavirin were fatigue, headache, nausea, insomnia and anemia.<sup>27</sup>

#### Ribavirin

The hemolytic anemia associated with ribavirin therapy may result in worsening of cardiac disease that has led to fatal and nonfatal myocardial infarctions. Significant teratogenic and embryocidal effects have been demonstrated in all animal species exposed to ribavirin. Therefore, ribavirin therapy is contraindicated in women who are pregnant and in the male partners of women who are pregnant.<sup>28</sup>

### Mavyret

In subjects receiving G/P for 8, 12, or 16 weeks, the most commonly reported adverse reactions of all intensity % were headache, fatigue and nausea.<sup>29</sup>

#### **Epclusa**

The most common adverse reactions (incidence greater than or equal to 10%, all grades) observed with treatment with Epclusa for 12 weeks are headache and fatigue. The most common adverse reactions (incidence

greater than or equal to 10%, all grades) observed with treatment with Epclusa and ribavirin for 12 weeks in patients with decompensated cirrhosis are fatigue, anemia, nausea, headache, insomnia and diarrhea.

### 12.12.5. Risks of Developing HCV

The risks of chronic HCV include severe acute inflammation of the liver that could lead to liver failure requiring a liver transplant. HCV may also cause a severe type of acute infection called fibrosing cholestatic HCV, that can cause severe liver injury, jaundice (yellowing of the eyes and skin), and progressive liver dysfunction.

#### 12.13. Risk of HCV Transmission

There is a small risk of transmission of HCV from the study subject to intimate partners during sexual activity. This risk is very low and should be reduced even further due to requirements for subjects to use barrier protection during sexual activity.

#### 12.14. Potential Benefits

The results from the study could be applied in the future to subjects (including those in the study) who stand to benefit from the information. Subjects will experience clinical benefits as their kidney function and quality of life should vastly improve following transplant. The study involves the risks of phlebotomy, echocardiography, Fibroscan, development of chronic HCV, and loss of confidentiality, but there is a potential for future benefit for both subjects in the study and for future subjects, the risk/benefit ratio is favorable.

#### 12.15. Alternatives

The use of the medications for this study requires that certain other medications not be used. Therefore, the alternative is to not participate in this study and to continue having the option to take these medications.

#### 12.16. Ethical Considerations

The main ethical considerations in this trial are non-maleficence, respect for persons, and autonomy. Our selection criteria are designed to select subjects who are at substantial risk of death and health complications because of end-stage renal disease and chronic dialysis treatment. Transplantation with a HCV-positive kidney and then treatment for HCV also involve risks, but it is plausible that survival and quality of life will still improve after transplantation compared to the alternative of multiple additional years on dialysis. Our informed consent procedures are designed to enable individuals to make decisions that are consistent with their values. We will enumerate the many possible risks and plausible benefits. The processes of informed consent in this study will be conducted so that patients can ask questions, confer with their primary nephrologists and develop a full understanding of the trial procedures and risks, all of which is consistent with respect for persons. Lastly, subjects in the trial will retain the ability to consider organ offers and decide whether to accept an organ based on their own judgment about the value of that particular organ and after getting advice from their transplant team.

## 13 CHAPTER 11: GOOD CLINICAL PRACTICE

This study is to be conducted accordance with applicable US government regulations and international standards of Good Clinical Practice, University of Pennsylvania requirements, and applicable institutional research policies and procedures.

This protocol and any amendments will be submitted to the FDA and a properly constituted IRB in agreement with local legal prescriptions for formal approval of the study conduct. The principal investigators will not commence the study until the IRB has issued written approval to the PIs.

All subjects for this study will be provided a consent form describing this study and providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the IRB for the study. The formal consent of a subject, using the IRB-approved consent form, must be obtained before that subject undergoes any study procedure. The consent form must be signed by the subject or legally acceptable surrogate, and the investigator-designated research professional obtaining the consent.

## 14 CHAPTER 12: REFERENCES

- 1. Sulkowski M, Hezode C, Gerstoft J, et al. Efficacy and safety of 8 weeks versus 12 weeks of treatment with grazoprevir (MK-5172) and elbasvir (MK-8742) with or without ribavirin in patients with hepatitis C virus genotype 1 mono-infection and HIV/hepatitis C virus co-infection (C-WORTHY): a randomised, open-label phase 2 trial. *Lancet*. 2015;385(9973):1087-1097.
- Lawitz E, Gane E, Pearlman B, et al. Efficacy and safety of 12 weeks versus 18 weeks of treatment with grazoprevir (MK-5172) and elbasvir (MK-8742) with or without ribavirin for hepatitis C virus genotype 1 infection in previously untreated patients with cirrhosis and patients with previous null response with or without cirrhosis (C-WORTHY): a randomised, open-label phase 2 trial. *Lancet*. 2015;385(9973):1075-1086.
- 3. Forns X, Gordon SC, Zuckerman E, et al. Grazoprevir and elbasvir plus ribavirin for chronic HCV genotype-1 infection after failure of combination therapy containing a direct-acting antiviral agent. *Journal of hepatology.* 2015;63(3):564-572.
- 4. Zeuzem S, Ghalib R, Reddy KR, et al. Grazoprevir-Elbasvir Combination Therapy for Treatment-Naive Cirrhotic and Noncirrhotic Patients With Chronic Hepatitis C Virus Genotype 1, 4, or 6 Infection: A Randomized Trial. *Annals of internal medicine*. 2015;163(1):1-13.
- 5. Reese PP, Abt PL, Blumberg EA, Goldberg DS. Transplanting Hepatitis C-Positive Kidneys. *The New England journal of medicine*. 2015;373(4):303-305.
- 6. O'Leary JG, Neri MA, Trotter JF, Davis GL, Klintmalm GB. Utilization of hepatitis C antibody-positive livers: genotype dominance is virally determined. *Transpl Int.* 2012;25(8):825-829.
- 7. Reddy KR FS, et al. Ledipasvir/Sofosbuvir with Ribavirin for the Treatment of HCV in Patients with Post Transplant Recurrence: Preliminary Results of a Prospective, Multicenter Study. *Hepatology*. 2014;60:200A.
- 8. Reese PP, Abt PL, Blumberg EA, et al. Twelve-Month Outcomes After Transplant of Hepatitis C-Infected Kidneys Into Uninfected Recipients: A Single-Group Trial. *Ann Intern Med.* 2018;169(5):273-281.
- 9. McLean RC, Reese PP, Acker M, et al. Transplanting hepatitis C virus-infected hearts into uninfected recipients: A single-arm trial. *Am J Transplant*. 2019;19(9):2533-2542.
- 10. Roth D ND, Bruchfeld A, et al. C-Surfer: Grazoprevir Plus Elbasvir In Treatment-Naïve and Treatment-Experienced Patients with Hepatitis C Virus Genotype 1 Infection and Chronic Kidney Disease. EASL 2015; 2015; Vienna, Austria.
- 11. Forns X, Lee SS, Valdes J, et al. Glecaprevir plus pibrentasvir for chronic hepatitis C virus genotype 1, 2, 4, 5, or 6 infection in adults with compensated cirrhosis (EXPEDITION-1): a single-arm, open-label, multicentre phase 3 trial. *The Lancet Infectious diseases*. 2017;17(10):1062-1068.
- 12. Asselah T, Kowdley KV, Zadeikis N, et al. Efficacy of Glecaprevir/Pibrentasvir for 8 or 12 Weeks in Patients With Hepatitis C Virus Genotype 2, 4, 5, or 6 Infection Without Cirrhosis. *Clinical gastroenterology and hepatology: the official clinical practice journal of the American Gastroenterological Association.* 2018;16(3):417-426.
- 13. Gane E, Lawitz E, Pugatch D, et al. Glecaprevir and Pibrentasvir in Patients with HCV and Severe Renal Impairment. *The New England journal of medicine*. 2017;377(15):1448-1455.
- 14. Feld JJ, Jacobson IM, Hezode C, et al. Sofosbuvir and Velpatasvir for HCV Genotype 1, 2, 4, 5, and 6 Infection. *The New England journal of medicine*. 2015;373(27):2599-2607.
- 15. Foster GR, Afdhal N, Roberts SK, et al. Sofosbuvir and Velpatasvir for HCV Genotype 2 and 3 Infection. *The New England journal of medicine*. 2015;373(27):2608-2617.
- 16. Goldberg DS, Halpern SD, Reese PP. Deceased organ donation consent rates among racial and ethnic minorities and older potential donors. *Crit Care Med.* 2013;41(2):496-505.

- 17. Pawlak R RJ, Maranan G, Michel-Treil V, Schutzbank T. A Comparative Evaluation of the Siemens VERSANT HCV Genotype 2.0 (LiPA) and GenMark eSensor HCV Direct Genotyping Tests. CVS 2013 Covance; 2013.
- 18. Dahl A HD, Ogorek T, Hansen G. Comparison of the GenMark Direct Genotype Assay with the LiPA Genotype Assay Using a Diverse Spectrum of HCV Clinical Samples Encountered in a High Risk Inner City HCV Population. CVS 2013 Hennepin; 2013.
- 19. Woodberry M SK, Castor J, Cook L, Jerome K. Genotyping of Hepatitis C Virus by the Genmark DX Esensor HCVG Direct Test. CVS 2013 UW-Seattle 2013.
- 20. Quest Diagnostics, Inc. (December 2014). Test summary guide. Hepatitis C Viral RNA Genotype 1 NS5a Drug Resistance.
  <u>www.questdiagnostics.com/testcenter/testguide.action?dc=TS\_HCV\_NS5A\_Genotype&tabview=true</u>
  Accessed March 14, 2016.
- 21. Begovac J, Krznaric J, Bogdanic N, Mocibob L, Zekan S. Successful treatment of genotype 3 hepatitis C infection in a noncirrhotic HIV infected patient on chronic dialysis with the combination of sofosbuvir and velpatasvir: A case report. *Medicine (Baltimore)*. 2018;97(51):e13671.
- 22. Smolders EJ, de Kanter CT, van Hoek B, Arends JE, Drenth JP, Burger DM. Pharmacokinetics, Efficacy, and Safety of Hepatitis C Virus Drugs in Patients with Liver and/or Renal Impairment. *Drug Saf.* 2016;39(7):589-611.
- 23. Liu Q, Mittal R, Emami CN, Iversen C, Ford HR, Prasadarao NV. Human isolates of Cronobacter sakazakii bind efficiently to intestinal epithelial cells in vitro to induce monolayer permeability and apoptosis. *J Surg Res.* 2012;176(2):437-447.
- 24. Merck Sharp & Dohme Corporation (January 2016). ZEPATIER™ tablets. Highlights of Prescribing Information. 2016.
- 25. Merck Sharp & Dohme Corporation (July 2015). Elbasvir (MK-8742). Investigator's Brochure (8th Ed.). 2015.
- 26. Merck Sharp & Dohme Corporation (July 2015). Grazoprevir (MK-5172). Investigator's Brochure (10th Ed.). 2015.
- 27. Gilead Sciences, Inc. (August 2015). Sovaldi® (sofosbuvir) tablets. Highlights of Prescribing Information. 2015.
- 28. Sandoz, Inc. (May 2015) Ribavirin capsule. Highlights of Prescribing Information. 2015. http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=dc637c8f-9669-4bc5-8787-1fd5abaa588e.
- 29. Mavyret US Package Insert, AbbVie Inc., 2017. URL: <a href="http://www.rxabbvie.com/pdf/mavyret\_pi.pdf">http://www.rxabbvie.com/pdf/mavyret\_pi.pdf</a>. Accessed September 5 2019.